#### The GlaxoSmithKline group of companies

201973

| Division | : Worldwide Oncology Development |
|------------------|-------------------------------------|
| Information Type | : Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for a Phase I/II Dose Escalation and Expansion Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of GSK525762 in Combination with Fulvestrant in Subjects with Hormone Receptor-Positive/HER2-Negative (HR+/HER2-) Advanced or Metastatic Breast Cancer. |
|---|---|---|
| <b>Compound Number</b> | : | GSK525762 |
| Effective Date | : | 11-AUG-2020 |

### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Phase I Clinical Study Report for Protocol 201973. This includes the Primary Clinical Study Report (CSR) and any End-of-Study outputs that will be generated.
- This RAP is intended to describe the planned efficacy, safety and pharmacokinetics analyses required for Phase I of the study.
- This RAP will be provided to the study team members to convey the content of Phase I data review and interim analysis deliverables, as well as to provide details of the Statistical Analysis Complete (SAC) deliverable.

#### **RAP Author:**

| Author | Date |
|---|---|
| Senior Biostatistician, Biostatistics FSP, PAREXEL employee on behalf of GlaxoSmithKline | 30-JUL-2020 |

Copyright 2020 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

### The GlaxoSmithKline group of companies

201973

# **RAP Team Reviewers:**

| Reviewer | Date | Approval Method |
|---|---|---|
| Clinical Scientist, Oncology Clinical Development | 10-AUG-2020 | Email |
| Director, Clinical Pharmacology Modelling and Simulation, GSK | 03-AUG-2020 | Email |
| Medical Director, Oncology Clinical Development | 07-AUG-2020 | Email |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Senior Statistics Director, Biostatistics, GSK | 11-AUG-2020 | Email |
| PPD Programming Director, Biostatistics, GSK | 31-JUL-2020 | Email |

201973

# TABLE OF CONTENTS

| | | PAGE |
|---|---|---|
| RA | P AUTHOR: | 1 |
| RA | P TEAM REVIEWERS: | 2 |
| CLI | INICAL STATISTICS AND CLINICAL PROGRAMMING LINE APPROVALS: | 2 |
| 1. | INTRODUCTION | 6 |
| 2. | SUMMARY OF KEY PROTOCOL INFORMATION 2.1. Changes to the Protocol Defined Statistical Analysis Plan 2.2. Study Objective(s) and Endpoint(s) | 6<br>6 |
| | 2.4.1. Dose Escalation Phase | 11 |
| 3. | PLANNED ANALYSES 3.1. Interim Analyses 3.1.1. Dose Escalation Phase 3.1.2. Dose Expansion Phase 3.1.2.1 Interim Futility Analysis 3.1.2.2 Interim Efficacy Analyses 3.1.2.3 Displays to be Created for Dose Expansion Review 3.2. Final Analysis | 12<br>13<br>14<br>14<br>16 |
| 4. | ANALYSIS POPULATIONS | |
| 5. | CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS 5.1. Study Treatment and Sub-group Display Descriptors 5.2. Reporting Conventions 5.3. Baseline and Post-Baseline Definitions 5.3.1. Change from baseline 5.3.2. Multiple Assessments 5.4. Multicentre Studies 5.5. Examination of Covariates, Other Strata, and Subgroups 5.5.1. Covariates and Other Strata 5.5.2. Examination of Subgroups 5.6. Other Considerations for Data Analyses and Data Handling Conventions | 20<br>21<br>22<br>23<br>23<br>23<br>23 |
| 6. | STUDY POPULATION ANALYSES 6.1. Overview of Planned Study Population Analyses 6.2. Disposition of Subjects 6.3. Protocol Deviations 6.4. Demographic and Baseline Characteristics 6.5. Concomitant Medications | 24<br>24<br>25 |

201973

7.1. 7.2. Summary Measures 28 7.3. 7.4. 8.2. 8.3. Adverse Events Leading to Discontinuation of Study Treatment and 8.4. 8.5. 8.6. 8.7. 8.8.1. 8.8.5. Liver Events 38 9.1.1.1. 9.1.1.2. 9.1.2. Summary Measure .......40 10. PHARMACODYNAMIC ANALYSIS.......40 11. OTHER STATISTICAL ANALYSES .......40 11.1. Value Evidence and Outcomes.......40 Appendix 1: Protocol Deviation Management and Definitions for Per Appendix 2: Schedule of Activities .......43 Appendix 3: Assessment Windows .......44 Appendix 4: Study Phases and Treatment Emergent Adverse 13.4. Events 45 Treatment States for Disease Response Data .......45 13.5. Appendix 5: Data Display Standards & Handling Conventions..................47 

201973

13.7.1. Premature Withdrawals......58 13.9. Appendix 9: Population Pharmacokinetic (PopPK) Analyses .......64 13.10.1. Abbreviations ......65 13.10.2. 13.11. Appendix 11: List of Data Displays......67 Data Display Numbering .......67 13.11.1. Mock Example Shell Referencing .......67 13.11.2. 13.11.3. Deliverables 67 13.11.4. Efficacy Tables .......70 13.11.5. Efficacy Figures ......71 13.11.6. 13.11.7. Safety Tables ......72 Pharmacokinetic Tables.....81 13.11.8. 13.11.9. Pharmacokinetic figures......83 ICH Listings ......84 13.11.10. Non-ICH Listings. 90 13.11.11. 13.12. Appendix 12: Example Mock Shells for Data Displays .......93

201973

### 1. INTRODUCTION

The purpose of this RAP is to describe the analyses to be performed in support of the Clinical Study Report for GSK Protocol 201973.

| Revision Chronology: | | |
|----------------------|-------------|----------------|
| Original | 11-AUG-2016 | 2015N238773_00 |
| Amendment No. 1 | 21-OCT-2016 | 2015N238773_01 |
| Amendment No. 2 | 31-JAN2017 | 2015N238773_02 |
| Amendment No. 3 | 07-MAR-2017 | 2015N238773_03 |
| Amendment No. 4 | 18-OCT-2017 | 2015N238773_04 |
| Amendment No. 5 | 11-SEP-2018 | 2015N238773_05 |
| Amendment No. 6 | 06-MAY-2020 | 2015N238773_06 |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There are no changes to the protocol defined statistical analysis as per the latest protocol amendment.

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To determine a recommended Phase 2 dose (RP2D) of GSK525752, when given in combination with fulvestrant, in women with advanced or metastatic hormone receptor-positive/HER2-negative breast cancer (HR+/HER2-BC). | Safety profile (e.g., adverse events [AEs], serious adverse events [SAEs], dose-limiting toxicities [DLTs], dose reductions or delays), overall response rate (ORR; defined as complete response [CR] rate plus partial response [PR] rate), pharmacokinetic (PK) parameters. |
| Secondary Objectives | Secondary Endpoints |
| To determine the safety, tolerability and maximum tolerated dose (MTD) of GSK525762, when given in combination with fulvestrant in women with advanced or metastatic HR+/HER2-BC. | AEs, SAEs, dose reductions or delays, withdrawals due to toxicities and changes in safety assessments (e.g., laboratory parameters, vital signs, electrocardiogram [ECG], cardiotoxicity, gastrointestinal, etc.). |
| To evaluate clinical activity of<br>GSK525762 and fulvestrant, when given<br>in combination, in women with advanced<br>or metastatic HR+/HER2-BC. | Disease control rate (DCR; defined as rate of CR plus PR plus stable disease [SD]), duration of response (DoR), and progression-free survival (PFS). |

201973

| Objectives | Endpoints |
|---|---|
| To characterize the exposure to GSK525762 and fulvestrant, when given in combination, in women with advanced or metastatic HR+/HER2-BC. | Concentrations of GSK525762, GSK525762 relevant metabolites, and fulvestrant following administration in combination. |
| <b>Exploratory Objectives</b> | Exploratory Endpoints |
| To evaluate additional measures of clinical activity of GSK525762 and fulvestrant, when given in combination, in women with advanced or metastatic HR+/HER2-BC. | Overall survival (OS). |
| To characterize the pharmacodynamics of GSK525762 and fulvestrant, when given in combination, in women with advanced or metastatic HR+/HER2-BC. | Transcriptomic and/or protein changes in<br>molecular markers of BET inhibition and<br>HR signalling in tumor tissue. (Analyses<br>may not be conducted if insufficient<br>sample size.) |
| To identify potential indicators of sensitivity or response to GSK525762 and fulvestrant, when given in combination, in women with advanced or metastatic HR+/HER2-BC. | <ul> <li>Mutational analysis of tumor tissue;<br/>correlation of baseline somatic and<br/>tumor-specific genetic and genomic<br/>profiles with response. (Analyses may<br/>not be conducted if insufficient sample<br/>size.)</li> </ul> |
| To describe the kinetics of tumor growth in the presence of GSK525762 and fulvestrant for each treatment and investigate the relationship between tumor growth kinetics and clinical activity. | Tumor size over time, tumor growth rate constants, and time to tumor growth, predicted by the model parameters defining relationships with clinical activity parameters. |
| To evaluate the exposure-response<br>relationship between GSK525762 and/or<br>fulvestrant exposure and safety and<br>efficacy parameters. | Relationship between GSK525762 and/or fulvestrant exposure markers (e.g., dose, C <sub>min</sub> , C <sub>max</sub> ), and safety and efficacy parameters. |
| To evaluate the effect of GSK525762 and fulvestrant, when given in combination, on symptoms and quality of life. | Change from baseline in EORTC-QLQ-<br>C30 and EORTC-QLQ-BR23<br>questionnaires. Changes from baseline in<br>select items from the PRO-CTCAE. |
| To evaluate ESR1 mutational status as a potential indicator of sensitivity and/or response to GSK525762 and fulvestrant, when given in combination, in women with advanced or metastatic HR+/HER2-BC. | Targeted sequencing to determine correlation between ESR1 mutations and clinical response. |

### 2.3. Study Design



#### Design Features

- Phase I of the study is designed as a parallel, single-arm, dose escalation/expansion phase to determine the RP2D based on safety, tolerability, PK and efficacy profiles observed after oral administration of GSK525762 in combination with fulvestrant, in advanced or metastatic HR+/HER2- BC subjects. The combination of GSK525762 plus fulvestrant will be evaluated in an open-label fashion in separate populations (i.e., cohorts) of subjects. Subjects will be enrolled into one of the following cohorts based on treatment history:
  - Cohort 1 Subjects with disease that relapsed during prior treatment or within 12 months after completing adjuvant therapy with an aromatase inhibitor (AI), or disease that progressed during prior treatment with an AI for advanced/metastatic disease. Prior ovarian suppression and/or tamoxifen are allowed, given all other criteria are met.
  - 2. <u>Cohort 2</u> Subjects with disease that progressed during prior treatment with the combination of a CDK4/6 inhibitor (e.g., palbociclib) plus letrozole for advanced/metastatic disease. Prior ovarian suppression and/or tamoxifen are allowed, given all other criteria are met.
- Phase I will follow a modified toxicity probability interval (mTPI) design, assuming (a) approximately 30 subjects will complete the DLT evaluation period and (b) the true underlying toxicity rate for GSK525762 in

201973

#### **Overview of Study Design and Key Features**

combination with fulvestrant falls within the range of 25% to 35%, centered at 30%.

- Cohort 1 may enrol up to 35 subjects, while Cohort 2 may enrol up to 32 subjects. However, the total number of subjects enrolled into each cohort may vary, as interim analyses for safety and efficacy may terminate enrolment within a cohort if the observed DLT rate exceeds the maximum permitted toxicity rate per the mTPI, or if the efficacy rate does not exceed the historical ORR.
- Dosing will begin at dose level 1 (DL1), with subjects administered GSK525762 at 60 mg orally once daily and fulvestrant at 500 mg intramuscularly (IM) on Days 1, 15 and 29 of Cycle 1 and then monthly thereafter. Subjects will be enrolled into cohorts based on their treatment history. Once three evaluable subjects (total, irrespective of cohort) have cleared the DLT evaluation period of 28 days, then an mTPI method will be used to determine whether to dose escalate to DL2 (if there is no DLT), reduce dose to DL-1 (if there are two or three DLTs), or continue enrolling subjects at DL1 (if there is one DLT). Up to 10 additional subjects may be enrolled in groups of approximately three at DL1 prior to a final dose escalation/de-escalation decision. If DL-1 is tested and found to be safe, then re-evaluation of DL1 may be attempted, if guided by the model. If both DL-1 and DL1 are being evaluated, then subjects will be randomized 1:1 to either DL-1 or DL1.
- Once a sentinel group of 3-10 evaluable subjects has cleared the DLT evaluation period of 28 days at DL1, the two cohorts will open at DL2. The DL2 DLT evaluation will occur as described for DL1, with a sentinel group of 3-10 evaluable subjects spread across the two cohorts.
- For each cohort, enrolment within the cohort may be stopped due to futility if the Bayesian predictive probability of confirmed response rate ≥25% (target) is small. Guidelines for interim futility analysis decision rules for the 10th through 34th evaluable subject are presented in Section 3.1.2.1, Interim Futility Analysis. The guidelines specify the number of subjects with confirmed responses needed for continued enrolment versus stopping for futility when the total sample size is <34 subjects in the cohort.
- The decision to proceed to Phase II will be based on the totality of data from Phase I, including safety, efficacy and PK data.
- While the overall study goals and design remain the same, changes have been made to Phase I of the study in order to address the emerging data and better define the patient population most likely to benefit from the combination treatment of GSK525762 plus fulvestrant. The following are to be noted:
  - 1. DL1 Cohort 1 (60 mg, AI failures) will enrol up to 35 subjects, as per Protocol Amendment 5.
  - 2. DL1 Cohort 2 (60 mg, CDK4/6 + AI failure) change in inclusion criteria and to the number of subjects to be enrolled is detailed below.

201973

| Overview of S | Study Design and Key Features |
|---|---|
| | 3. DL2 (80 mg) both cohorts (Cohort 1 and Cohort 2) – enrolment is closed based on decreased tolerability and lack of efficacy, as per protocol guidance. |
| | • Enrolment into DL1 (60mg) Cohort 2 is modified. Subjects previously treated with the combination of a CDK4/6 inhibitor (e.g., palbociclib) plus AI for advanced or metastatic disease will be enrolled as follows: |
| | <ul> <li>Up to 32 subjects with measurable disease who have progressed after<br/>greater than or equal to 12 months of prior treatment with CDK4/6<br/>inhibitor plus AI.</li> </ul> |
| | <ul> <li>Up to 16 subjects with bone only disease who have progressed after<br/>greater than or equal to 12 months of prior treatment with CDK4/6<br/>inhibitor plus AI.</li> </ul> |
| | <ul> <li>Prior ovarian suppression and/or tamoxifen will be allowed, given all<br/>other criteria are met.</li> </ul> |
| Dosing | The projected dose levels of GSK525762 for Phase I dose escalation are 60 mg (DL1) and 80 mg (DL2), each administered orally once daily. If unacceptable toxicity is observed at 60 mg, then 40 mg once daily may be explored (referred to as DL-1). |
| | The projected dose level of fulvestrant is the approved dose regimen of 500 mg IM on Days 1, 15 and 29 of Cycle 1 and then monthly thereafter. |
| Time and<br>Events | Refer to Tables 4 and 5 in Section 7.1 of the Protocol. |
| Treatment<br>Assignment | Study Phase I is an open label, single-arm phase. If one dose level is open for enrolment, subjects will be assigned to the dose at that level. If more than one dose level is open for enrolment, subjects will be randomly assigned to one of the open dose levels with 1:1 allocation. |
| Interim<br>Analysis | After at least 10 evaluable subjects become available in each expansion cohort, futility analyses will be performed. After that, interim analysis may be conducted after every 5 evaluable subjects become available. Phase I interim analyses may also be undertaken for each expansion cohort after the last subject enrolled in the cohort has been followed for 6 months or has progressed, died, or withdrawn from the study treatment. |
| | Enrolment to an individual cohort may be stopped due to futility if the Bayesian posterior probability that the confirmed ORR ≥25% in Cohort 1 (AI failure) or ≥20% in Cohort 2 (CDK4/6 + AI failure) is small (see Tables 1 and 2). Enrolment may also be stopped due to futility if the equivalent of no response is observed in the first 10 enrolled evaluable subjects in that cohort or if fewer than 2 confirmed responses are observed in the first 14 and 19 evaluable subjects in Cohort 1 and Cohort 2, respectively. |
| | Decision-making criteria for futility are presented in Table 9 for Cohort 1 (AI failure) and Table 10 for Cohort 2 (CDK4/6 + AI failure) in Section 9.3.2 of the Protocol. |
| Final<br>Analysis | The study will be considered complete for purposes of a final analysis when approximately 70% of all enrolled subjects have died. |

201973

| Overview | Overview of Study Design and Key Features |
|---|---|
| Study<br>Status | The totality of Phase I data assessed at the interim analysis does not support continuing investigation of GSK525762 (molibresib) in combination with fulvestrant for the treatment of HR+/HER2- advanced or metastatic breast cancer patients. As interim data failed to demonstrate meaningful clinical benefit in this patient population, enrolment into the study is now closed and the study will not incorporate Phase II. |
| | With the implementation of Amendment 06, specific assessments and collection of survival follow-up data will no longer be required. The study will conclude when the last subject has completed/discontinued study treatment and completed the end of treatment visit. |

### 2.4. Statistical Hypotheses / Statistical Analyses

#### 2.4.1. Dose Escalation Phase

Dose escalation decisions will be based on the totality of clinical safety assessment data, as well as PK data. All analyses will be descriptive in nature.

### 2.4.2. Dose Expansion Phase

For evaluation of efficacy in Cohort 1 (AI Failure) in Phase I, the primary goal is to demonstrate a clinically meaningful response rate, defined as an ORR (equal to CR rate + PR rate) of 25% relative to a 10% response rate suggesting no activity. This will be achieved by testing the null hypothesis of  $P0 \le 0.1$  versus the alternative of P1 > 0.25, assuming the maximum response rate for an ineffective drug is 10% and the minimum response rate for an effective drug is 25%.

For evaluation of efficacy in Cohort 2 (CDK4/6 + AI Failure) in Phase I, the primary goal is to demonstrate a clinically meaningful response rate in subjects with measurable disease only. In this cohort, a meaningful response rate is defined as an ORR of 20% relative to a 5% response rate suggesting no activity. This will be achieved by testing the null hypothesis of  $P0 \le 0.05$  versus the alternative of P1 > 0.20, assuming the maximum response rate for an ineffective drug is 5% and the minimum response rate for an effective drug is 20%.

Bayesian statistics will be employed to calculate the posterior probability that the ORR  $\geq$ 25% and  $\geq$ 10% for Cohort 1 (AI Failure) and  $\geq$ 20% and  $\geq$ 5% for Cohort 2 (CDK4/6+AI Failure) at interim assuming a Beta prior for the Binomial distributed data. A weak prior Beta (0.0125, 0.0875) for Cohort 1 and (0.005, 0.095) for Cohort 2 will be used, which is equivalent to the information present in 0.1 subjects.

201973

#### 3. PLANNED ANALYSES

### 3.1. Interim Analyses

#### 3.1.1. Dose Escalation Phase

No formal interim analysis will be performed for dose escalation decisions in Phase I. These decisions instead will be based primarily on ongoing data review using Spotfire visualization, with additional outputs created by Statistics and Programming if necessary. The assessments driving dose escalation decisions will focus on the safety and tolerability of GSK525762 combined with fulvestrant within each combination of dose level x cohort. Descriptive analyses will be based on the All Treated Population (defined in Section 4, Analysis Populations).

The mTPI design rules, together with predicted dose-limiting toxicity rates at all dose levels, will support the determination of whether to move forward with dose escalation and expansion as planned for Phase I. The mTPI design rests on the assumptions that (a) approximately 30 subjects will complete the DLT evaluation period and (b) the true underlying toxicity rate for GSK525762 in combination with fulvestrant falls within the range of 25% to 35%, centred at 30%.

The monitoring rules guiding dose escalation are provided in Figure 1, below. Columns provide the numbers of subjects treated at the current dose level, while rows provide the corresponding numbers of subjects experiencing toxicity. Entries within the table represent the dose-finding decisions of escalating the dose (E), staying at the same dose (S), and de-escalating the dose (D). If the current dose is at the highest dose level and the decision is E, then the highest dose level is below MTD and the next subject(s) will be treated at the same dose level. In addition, decision U indicates that the current dose level is of unacceptably high toxicity and should be subsequently excluded from the trial. For example, when one of three subject experiences toxicity, the decision is located at row 1/column 3, which is to stay at current dose level (S). Consequently, the next cohort of subjects will be treated at the same dose level currently being used. If none of three subjects experience toxicity, the decision is shown at row 0/column 3, which is to escalate (E) to a higher dose (if available) or to otherwise stop dose escalation when 6 evaluable subjects have been treated at the current dose. Thus, the next cohort of subjects may be treated at the next higher dose level. If three of three subjects experience toxicity, the decision is to de-escalate (DU) to the next lower dose level and subsequently exclude the current dose from the trial, because the high toxicity level is unacceptable.

201973

Figure 1 – Modified toxicity probability interval (mTPI) method dose finding rules



The spreadsheet was generated based on a beta/binomial model and precalculated before trial initiation. The letters in different colors are computed based on the decision rules under the mTPI method and represent different dose-finding actions. In addition to actions de-escalate the dose (D), stay at the same dose (S), and escalate the dose (E), the table includes action unacceptable toxicity (U), which is defined as the execution of the dose-exclusion rule in mTPI.

# 3.1.1.1. Displays to be Created for Dose Escalation Review

Review of preliminary data will be performed after 3-10 evaluable subjects complete the DLT evaluation period of 28 days for each dosing level.

For the first dose escalation meeting, spreadsheets containing relevant study data will be supplied by the study data manager. For dose escalation meetings after the first cohort, SDTM datasets will be uploaded and made available in Spotfire. Both GSK and PAREXEL personnel will have access to Spotfire and will be able to view subject-level data. In addition to the review of Spotfire data visualisations, summary displays may be provided by Statistics and Programming, as necessary.

GSK has in place a comprehensive and robust review process of all data. During the dose expansion cohorts, all safety, efficacy, and PK data emerging from the study will be reviewed by a Joint Team comprised of participating investigators and study coordinators, together with staff involved in the conduct of the study (i.e. Medical Monitor, Program Lead Physician, Safety (Pharmacovigilance) Physician, Clinical Pharmacokineticist, Statistician, and Clinical Scientist).

Furthermore, multiple review points and mechanisms will be implemented to safeguard subject safety during the conduct of Phase I. The key elements of such safety reviews will include regularly scheduled data reviews and investigator meetings, specific safety

201973

review meetings, and a comprehensive dose selection meeting to be held at the end of Phase I.

Prior to determining a dose level for the next cohort, exploratory analyses may be conducted to assess the potential relationships between dose level and safety, PK, and pharmacodynamic parameters using all data from available cohorts.

The GSK study team, in collaboration with study investigators, will review all relevant data (as well as the results of any exploratory analyses) to determine whether the current dose showed acceptable toxicity and to decide the next dose level to be administered based on the totality of the data.

### 3.1.2. Dose Expansion Phase

### 3.1.2.1. Interim Futility Analysis

Interim data will be evaluated to monitor efficacy and safety, and a planned interim analysis will be performed when at least 10 evaluable subjects have been enrolled into each of the expansion cohorts at each DL. Enrolment may be stopped early in any of the expansion cohorts for toxicity or lack of efficacy. The decision criteria for early stopping for futility is based on the Bayesian Hierarchical model described below. The decision will be made for each individual prior treatment history-specific cohort.

For the futility interim analyses in each cohort, the enrolment for that cohort may be stopped due to futility if the posterior probability that the confirmed ORR ≥25% or ORR ≥20% in Cohort 1 and Cohort 2, respectively, is small (e.g., less than a 4% chance for a total sample size of 35 subjects). Enrolment may also be stopped due to futility if the equivalent of no objective response (i.e., no confirmed CR or PR) is observed in the first 10 evaluable subjects in that cohort or if fewer than 2 objective responses are observed in the first 14 and 19 evaluable subjects in Cohort 1 and Cohort 2, respectively. An evaluable subject is defined as a subject who has progressed, died, or withdrawn from the study treatment, or is still undergoing treatment and has completed at least two post-baseline disease assessments. For example, if 14 evaluable subjects show only one response at the time of interim analysis, then the cohort may be stopped for futility. Otherwise, enrolment within the respective cohort will continue to the target sample size.

Futility interim analysis decision rules for the 10th through 34th evaluable subject in Cohort 1 (AI Failure) and 10th through 31st evaluable subject in Cohort 2 (CDK4/6 + AI Failure) are presented in Tables 1 and 2, respectively. These rules, which are intended to function as guidelines, specify the number of objective responses (i.e., confirmed CRs or PRs) required to continue enrolment (vs. stop for futility) when the total target sample sizes are up to 35 in Cohort 1 and 32 in Cohort 2. Importantly, actual decisions will depend on the totality of the data.

201973

Table 1 – Decision Making Criteria for Assessing Futility in Cohort 1 (Al Failure)

| Number of Evaluable Subjects | ≤ This Number of Confirmed Responses to Stop Early for Futility | Probability of continuing enrolling when ORR=0.1 | Probability of continuing enrolling when ORR=0.25 |
|---|---|---|---|
| 10 | 0 | 0.6513 | 0.9437 |
| 11 | 0 | 0.6513 | 0.9437 |
| 12 | 0 | 0.6513 | 0.9437 |
| 13 | 0 | 0.6513 | 0.9437 |
| 14 | 1 | 0.3971 | 0.8843 |
| 15 | 1 | 0.3971 | 0.8843 |
| 16 | 1 | 0.3971 | 0.8843 |
| 17 | 1 | 0.3971 | 0.8843 |
| 18 | 1 | 0.3971 | 0.8843 |
| 19 | 1 | 0.3971 | 0.8843 |
| 20 | 1 | 0.3971 | 0.8843 |
| 21 | 2 | 0.2938 | 0.8674 |
| 22 | 2 | 0.2938 | 0.8674 |
| 23 | 2 | 0.2938 | 0.8674 |
| 24 | 2 | 0.2938 | 0.8674 |
| 25 | 2 | 0.2938 | 0.8674 |
| 26 | 2 | 0.2938 | 0.8674 |
| 27 | 3 | 0.2108 | 0.8511 |
| 28 | 3 | 0.2108 | 0.8511 |
| 29 | 3 | 0.2108 | 0.8511 |
| 30 | 3 | 0.2108 | 0.8511 |
| 31 | 3 | 0.2108 | 0.8511 |
| 32 | 4 | 0.1509 | 0.8369 |
| 33 | 4 | 0.1509 | 0.8369 |
| 34 | 4 | 0.1509 | 0.8369 |

201973

Table 2 – Decision Making Criteria for Assessing Futility in Cohort 2 (CDK4/6 + Al Failure)

| Number of Evaluable Subjects | ≤ This Number of<br>Confirmed Responses to<br>Stop Early for Futility | Probability of continuing enrolling when ORR=0.05 | Probability of continuing enrolling when ORR=0.2 |
|---|---|---|---|
| 10 | 0 | 0.4013 | 0.8926 |
| 11 | 0 | 0.4013 | 0.8926 |
| 12 | 0 | 0.4013 | 0.8926 |
| 13 | 0 | 0.4013 | 0.8926 |
| 14 | 0 | 0.4013 | 0.8926 |
| <u>15</u> | 0 | 0.4013 | 0.8926 |
| <u>16</u> | 0 | 0.4013 | 0.8926 |
| 17 | 0 | 0.4013 | 0.8926 |
| 18 | 0 | 0.4013 | 0.8926 |
| 19 | 1 | 0.2027 | 0.8566 |
| 20 | 1 | 0.2027 | 0.8566 |
| 21 | 1 | 0.2027 | 0.8566 |
| 22 | 1 | 0.2027 | 0.8566 |
| 23 | 1 | 0.2027 | 0.8566 |
| 24 | 1 | 0.2027 | 0.8566 |
| 25 | 1 | 0.2027 | 0.8566 |
| 26 | 1 | 0.2027 | 0.8566 |
| 27 | 2 | 0.1090 | 0.8362 |
| 28 | 2 | 0.1090 | 0.8362 |
| 29 | 2 | 0.1090 | 0.8362 |
| 30 | 2 | 0.1090 | 0.8362 |
| 31 | 2 | 0.1090 | 0.8362 |

### 3.1.2.2. Interim Efficacy Analyses

Interim efficacy analyses may also be performed for each expansion cohort after the last subject enrolled in the cohort has been followed for 6 months or has progressed, died, or withdrawn from the study treatment.

# 3.1.2.3. Displays to be Created for Dose Expansion Review

The All Evaluable Population (see Section 4, Analysis Populations) will be used for futility analyses. As subjects enrol at different times, not all subjects may be on study long enough to undergo multiple or even single post-baseline disease assessment(s). An evaluable subject is a subject who has progressed, died, or withdrawn from the study treatment, or is still undergoing treatment and has completed at least two post-baseline disease assessments.

The All Treated Population (see Section 4, Analysis Populations) will be used to produce study population, efficacy (other than futility), and safety summaries.

201973

The ORR is defined as the percentage of subjects in the population who show a best overall response (BOR) of confirmed CR or PR per RECIST v1.1. The ORR will be provided with its exact 95% confidence interval (CI). Subjects with unknown or missing response will be treated as non-responders (i.e., these subjects will be included in the denominator when calculating the percentage).

A listing of subject status and BOR will be provided. This listing will be sorted by date of the subject's first dose and will show whether each subject is still undergoing study treatment, whether the subject has had at least two post-baseline radiological disease assessments, whether the subject is considered evaluable for the futility analysis, and the subject's BOR (including confirmed and unconfirmed response).

Summaries, as well as data listings, of AEs, drug related AEs, AEs leading to study treatment discontinuation and other dose modifications, SAEs, fatal SAEs, study treatment related SAEs, exposure to GSK525762 and fulvestrant, and GSK525762 and fulvestrant dose modification(s) will be provided. In addition, summaries of laboratory assessments, vital signs, ECGs, Eastern Cooperative Oncology Group (ECOG) scores, and left ventricular ejection fraction (LVEF) results will be provided.

PK analysis will be performed using the PK Population (as defined in Section 4, Analysis Populations), with results presented by subgroups representing combinations of dose level x cohort, for GSK525762, its relevant metabolites, and fulvestrant (see Section 5.5.2 for subgroup descriptions). For further evaluation of the PK of GSK525762, the results within this study may also be compared to the results of other studies, wherein higher dose level(s) were administered.

Refer to Appendix 11: List of Data Displays for the full list of displays.

### 3.2. Final Analysis

The final analysis will be performed when approximately 70% of all enrolled subjects have died. Also, the final analysis will occur after all required database cleaning activities have been completed and both final database release (DBR) and database freeze (DBF) have been declared by Data Management.

As the study and project have been terminated, the primary analysis will occur once the termination decision has been confirmed, and the final analysis will occur once all ongoing subjects have completed the study.

As final analysis may be performed when some subjects are still in follow-up and additional data may be available by study closure, an amendement to this RAP may be performed, if needed for guiding a re-run of the analysis described below.

201973

### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Screened<br>Population | Subjects who consent to participate in the trial. | <ul><li> Screen failures</li><li> Enrolled subjects</li></ul> |
| All Treated<br>Population | Subjects who receive at least one dose of study treatment (GSK525762 or fulvestrant). In addition to primary analyses of study population, safety, and efficacy, this population will be used for decision-making during dose escalation. | <ul> <li>Study population</li> <li>Anti-cancer activity</li> <li>Safety</li> </ul> |
| Modified All<br>Treated<br>Population | All subjects who receive at least one dose of GSK525762 and fulvestrant. | <ul> <li>Efficacy</li> <li>Safety (if<br/>different from the<br/>All Treated<br/>population)</li> </ul> |
| All Evaluable<br>Population | Subjects who have at least two post-baseline radiological disease assessments or have progressed or died or permanently withdrawn from the study treatment. This population will be used for decision-making at the interim futility analysis. | <ul> <li>Dose escalation phase</li> <li>Interim futility analyses</li> </ul> |
| PK Population | Subjects from the All Treated Population for whom a PK sample is obtained and analysed. | PK analysis |

**NOTE:** Please refer to List of Data Displays, which details the population to be used for each display being generated.

#### 4.1. Protocol Deviations

Major protocol deviations (e.g., deviations related to study inclusion/exclusion criteria, conduct of the trial, subject management, or subject assessment) will be summarised and all protocol deviations will be listed.

Protocol deviations will be tracked by the study team throughout the study in accordance with the Protocol Deviation Specifications developed by PAREXEL. To ensure that all important deviations are captured and categorised in the protocol deviations dataset, data will be reviewed prior to DBF at the end of Phase I. This dataset will be the basis for all summaries and listings of protocol deviations, including a separate summary and separate listing dedicated to all deviations related to inclusion/exclusion criteria. These latter data displays will be based on data recorded on the inclusion/exclusion electronic case report form (eCRF).

201973 | Statistical Analysis Plan Statistical Analysis Plan for 201973 11 Aug 2020 | TMF-11735671 | 1.0

### **CONFIDENTIAL**

201973

As no Per Protocol Population has been defined for this study, protocol deviations will not be used to determine membership in any particular analysis population.

201973

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Data will be summarised and listed according to GSK reporting standards, as applicable. Summaries and listings will be displayed by or will otherwise incorporate the subgroups described below and in Section 5.5.2, Examination of Subgroups.

### 5.1. Study Treatment and Sub-group Display Descriptors

Data will be summarised and listed according to GSK reporting standards, as applicable. All data displays (tables, figures, and listings) will use the term "Subject" which reflects Clinical Data Interchange Standards Consortium (CDISC) and GSK Data Display Standards terminology. Tables, figures, and listings will be displayed by study treatment dose level. Actual dose levels will depend on outcomes of the dose escalation phase but will follow the same format. Subgroups described in Section 5.5.2, Examination of Subgroups, may also be used in summaries.

| <b>Treatment Description</b> | Treatment Label / Column<br>Header | Order <sup>[1]</sup> |
|---|---|---|
| GSK525762 60mg + fulvestrant 500 mg | GSK762 60 mg + FUL 500 mg | 1 |
| GSK525762 80mg + fulvestrant 500 mg | GSK762 80 mg + FUL 500 mg | 2 |
| Fulvestrant 500 mg | Fulvestrant 500 mg [2] | 3 |
| GSK525762 60mg | GSK762 60 mg <sup>[2]</sup> | 4 |
| GSK525762 80mg | GSK762 80 mg <sup>[2]</sup> | 5 |

#### **NOTES:**

- 1. Order represents treatments being presented in TFL, as appropriate.
- 2. Required only for tables that are displayed separately for individual treatment.

| Sub-Gr | Sub-Group Descriptions | | |
|---|---|---|---|
| Interac | active response technology (IRT) Data Displays for Reporting | | |
| Code | Description | Description [1] | Order [2] |
| A | DL1_COHORT1 | GSK762 60 mg + FUL 500mg<br>(AI Failure) | 1 |
| A | DL1_COHORT2 | GSK762 60 mg + FUL 500mg<br>(CDK4/6 + AI Failure < 12M) | 2 |
| A | DL1_COHORT2 | GSK762 60 mg + FUL 500mg<br>(CDK4/6 + AI Failure >= 12M) | 3 |

201973

| Sub-Gr | Sub-Group Descriptions | | |
|---|---|---|---|
| Interact | tive response technology (IRT) | <b>Data Displays for Reporting</b> | |
| Code | Description | Description [1] | Order [2] |
| A | DL1_COHORT2 | GSK762 60 mg + FUL 500mg<br>(CDK4/6 + AI Failure >= 12M<br>Bone Only Disease) | 4 |
| В | DL2_COHORT1 | GSK762 80 mg + FUL 500mg<br>(AI Failure) | 5 |
| В | DL2_COHORT2 | GSK762 80 mg + FUL 500mg<br>(CDK4/6 + AI Failure) | 6 |

#### NOTES:

- 1. The duration of 12 months equals, on average, 365.25 days.
- 2. Order represents the order of treatments as presented in each TFL display.

### 5.2. Reporting Conventions

- Unless otherwise specified, the denominator used in the calculation of percentages will be based on the number of subjects with non-missing values for the given scheduled visit and assessment or parameter.
- All data are reported according to the dose/regimen initially received by the subject.
- At minimum, data will be listed by treatment group, centre ID, and subject ID.
- Planned times relative to investigational product dosing will be used in all summary tables and figures, unless otherwise specified.
- Unscheduled visits will be included in the listing using actual time and will be used in deriving the maximum or minimum value over time (e.g. worst-case value post dose). However, unscheduled visits will not be included in summaries by planned time.
- Actual, rather than planned, sampling times will be used in the derivation of PK parameters and in the individual concentration-time plots. Planned times will be used in the descriptive summaries and mean/median plots. Listings of PK concentration-time data will be displayed by actual sampling times relative to dosing time.
- No formal assessment windows will be defined for the purpose of classifying measurements obtained outside of scheduled assessment times.
- Programmers should refer to GSK IDSL standards (as applicable) for decimal place conventions and expand if necessary. Unless stated otherwise, descriptive summaries will include n, mean, standard deviation (SD), median, minimum, and maximum for continuous variables and n and percentage for categorical variables. Minimum and maximum values will be displayed with the same precision as original source data, mean and median values will be displayed with one additional decimal place, and SD values will be displayed with two additional decimal places.

201973

- This is a multicentre study. Data from all study centres will be integrated into derivations and summaries without controlling for centre effects.
- Analyses will be performed using SAS statistical software version 9.4 or later. Programs will be imported into HARP, and the final outputs will be produced by running drivers in HARP. Some graphics may be produced using Tibco Spotfire Clinical Graphics, comprising S-Plus (R) version 7.0.6 or later.
- Deviations from any planned analyses in this RAP will be identified in the final CSR.

#### 5.3. Baseline and Post-Baseline Definitions

For all endpoints, baseline will be defined as the most recent (latest), non-missing assessment time-point prior to the first study treatment dose.

For enrolled subjects who do not receive the study treatment, baseline will be defined as the latest assessment time-point providing analysable data.

For laboratory data, baseline will be defined as the most recent, non-missing value from a central laboratory prior to the first study treatment dose. If there are no central labs collected for a subject, the most recent, non-missing value from a local laboratory prior to the first dose of study treatment will be defined as the baseline value.

For ECG analyses, the baseline value will be represented by the mean of the triplicate of the most recent (latest) assessment time-point prior to the first study treatment dose, if available. If Fridericia's QT Interval Corrected for Heart Rate (QTcF) results are not available at baseline, then the mean of the screening triplicate QTcF results will be used.

Unless otherwise stated, if baseline data are missing, then no derivations (e.g., change from baseline) will be performed and baseline will be set to missing.

### 5.3.1. Change from baseline

Following the initiation of treatment, absolute change from baseline will be calculated as: post-baseline value – baseline value.

Percent (i.e., relative) change from baseline will be calculated as: (absolute change from baseline value  $\div$  baseline value) x 100.

If either the baseline value or post-baseline value is missing, then both the absolute and relative changes from baseline will be set to missing.

# **5.3.2. Multiple Assessments**

All data will be reported as corresponding to a nominal visit, as no visit windows will be applied during dataset creation. Data from unscheduled visits will be included in summaries reporting worst-case post-baseline results only and in all relevant data listings.

For summaries in which data are collapsed across multiple planned time intervals, the means of intervals will be summarised.

201973

With the exceptions of ECG and echocardiogram (ECHO) or multiple gated acquisition (MUGA) assessments, if multiple assessments of the same type are performed on different days but reported for the same scheduled assessment, then only the worst-case assessment results for that scheduled assessment will be analysed.

With the exceptions of laboratory, ECG, and ECHO/MUGA assessments, the reporting of multiple assessments of the same type on the same date for the same visit or timepoint will be addressed by using the mean of the multiple reported measurements within analyses.

For laboratory assessments, data may be collected from both local and central laboratories for the same visit or timepoint, but, in such case, only data from the central laboratory will be analysed to maintain comparability across measurements and subjects.

For ECG and ECHO/MUGA assessments, both local investigator and central cardiologist readings will be performed for each visit/timepoint. For these assessments, only post-baseline data collected using the same method (i.e., ECG, ECHO vs. MUGA) and by the same source (i.e., local vs. central cardiologist read) as the baseline assessment will be used to derive change from baseline.

Data from all assessments, regardless of whether scheduled or unscheduled and performed singly or in multiple, will be included in the data listings.

#### 5.4. Multicentre Studies

Data from all participating centres will be pooled prior to analysis. It is anticipated that subject accrual will be spread thinly across centres and summaries of data by centre would be unlikely to be informative and will not, therefore, be provided.

### 5.5. Examination of Covariates, Other Strata, and Subgroups

#### 5.5.1. Covariates and Other Strata

No covariate-adjusted or stratified analyses are planned for this study.

# **5.5.2. Examination of Subgroups**

Subject subgroups to be included in analysis and reporting may be represented by (a) the study phases (Phase I vs. Phase II), (b) the combinations of dose level (e.g., DL-1, DL1, DL2) and cohort (Cohort 1 [AI Failure] vs. Cohort 2 [CDK4/6 + AI Failure]), and (c) the combinations of dose level, prior treatment, timing of a progressive disease response to prior treatment, and evidence of bone-only disease (see Section 5.1, Study Treatment and Sub-group Display Descriptors, for descriptions).

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined across multiple appendices:

201973

| Section | Component |
|---------|----------------------------------------------------------------|
| 13.3 | Appendix 3: Assessment Windows |
| 13.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 13.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 13.6 | Appendix 6: Derived and Transformed Data |
| 13.7 | Appendix 7: Reporting Standards for Missing Data |
| 13.8 | Appendix 8: Values of Potential Clinical Importance |

#### 6. STUDY POPULATION ANALYSES

### 6.1. Overview of Planned Study Population Analyses

Study population analyses will be based on the All Treated Population, unless otherwise specified. Analyses will include descriptive summaries and data listings of subject disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and treatment exposure, based on GSK Core Data Standards. Details of all planned displays are presented in Appendix 11: List of Data Displays.

### 6.2. Disposition of Subjects

Using the All Screened Population, the numbers and percentages of subjects in each analysis population (described in Section 4, Analysis Populations) will be summarised. A listing of subjects excluded from the analysis populations and both a summary and a listing of subject screening status and reasons for screen failure will be provided.

A summary of study treatment status will be provided. This display will show the number and percentage of subjects who are ongoing or discontinued study treatment and a summary of the primary reasons for discontinuation of study treatment. Reasons for study treatment discontinuation will be presented in the order that they are displayed on the eCRF. A listing of study treatment discontinuation will be generated. The listing will include last dose date, reasons for study treatment discontinuation, and study phase of discontinuation.

A summary of subject status and reason for study withdrawal will be provided. This display will show the number and percentage of subjects who either are ongoing or withdrew from the study. Primary reasons for study withdrawal will also be summarised. Reasons for study withdrawal will be presented in the order they are displayed in the eCRF. A listing of reasons for study withdrawal will also be included.

#### 6.3. Protocol Deviations

Only major protocol deviations will be summarised, whereas all protocol deviations (regardless of categorization) will be included in a listing. A separate listing dedicated to deviations related to inclusion/exclusion criteria will also be provided. Protocol deviations will be classified as "major" and "minor", based on Protocol Deviation Specifications.

201973

### 6.4. Demographic and Baseline Characteristics

Demographic and other baseline characteristics of subjects (e.g., age, race, ethnicity, sex, and body height and weight) will be both summarised and included in a listing. Age, height, and weight will be summarised as continuous variables, whereas sex, race, and ethnicity will be summarised as categorical variables. Age will be additionally summarised as a categorical variable using the EudraCT categories of 18-64, 65-84 and  $\geq$ 85 years and GSK IDSL categories of  $\leq$ 18, 18-65, and  $\geq$ 65 years. A separate listing dedicated to categorical age and both a separate summary and listing dedicated to race/racial combinations will also be provided.

Medical conditions present at screening will be separately summarised by past and current categories; both past and current conditions will be disclosed in a single listing. Medical conditions that are not pre-specified will be incorporated into the listing only.

Substance use, including history of smoking, tobacco, and alcohol, will be disclosed in a listing.

Disease characteristics at initial diagnosis and study screening will be summarised separately and provided in separate listings. As appropriate per summary, characteristics may include primary tumor type, stage, lesion status, time since initial diagnosis, and time since latest disease progression. Sites of metastatic disease at screening will be both summarised and included in a listing, and, lastly, a summary describing disease burden at baseline will be provided.

Anti-cancer therapy will be coded using the GSK drug coding dictionary. Separate summaries will be produced for prior anti-cancer therapy (dedicated to all therapies, including radiotherapies), prior dictionary-coded therapy, and number of therapy regimens. The details of prior and subsequent anti-cancer therapies will be disclosed in two listings, one for all therapies and one for radiotherapies. A summary of best response to the most recent prior anti-cancer therapy will also be provided.

Prior and on-treatment cancer-related surgical procedures will be summarized separately but included in the same listing.

#### 6.5. Concomitant Medications

Concomitant medications, coded using the GSK drug coding dictionary, will be both summarised and included in a listing. The summary will show the number and percentage of subjects taking concomitant medications by ingredient. Multi-ingredient products will be summarised by their separate ingredients rather than as a combination of ingredients. Anatomical-Therapeutic-Chemical (ATC) Level 1 (Body System) classification will be included in the created dataset but will not appear in the summary table or listing.

In the summary of concomitant medications, each subject will be counted once per unique ingredient. For example, if a subject takes Amoxycillin on two separate occasions, the subject is counted only once under the ingredient "Amoxycillin". In the summary of concomitant medications, the ingredients will be summarised by the base only. A single listing, incorporating both blood products and supportive care products, will be provided.

201973

Note that, in order to be considered a concomitant medication, the concomitant medication must have been taken at some point during the on-therapy window.

#### 7. EFFICACY ANALYSES

Efficacy analyses will be based on the Modified All Treated Population, unless otherwise specified. The results of all efficacy analyses will be presented by subject subgroup, defined by the combination of dose level, prior treatment, timing of a progressive disease response to prior treatment, and evidence of bone-only disease (see Section 5.5.2, Examination of Subgroups).

### 7.1. Endpoints / Variables

#### **Best Overall Response (BOR)**

BOR is defined as the best confirmed or unconfirmed response observed following the initiation of treatment through first documentation of progressive disease (PD) or initiation of new anti-cancer therapy, whichever occurs earlier. Responses following the onset of treatment will be assessed by the investigator per RECIST v1.1 criteria and, listed from best to worst, may include: CR, PR, SD (or non-CR/non-PD), PD, and not evaluable (NE).

#### **Objective Response Rate (ORR)**

ORR is defined as the percentage of subjects in the population who demonstrate a BOR of confirmed CR or PR, as assessed by the investigator per RECIST v1.1 criteria.

#### **Disease Control Rate (DCR)**

DCR is defined as the percentage of subjects in the population with a confirmed CR, confirmed PR, or SD lasting  $\geq 6$  months, as assessed by the investigator per RECIST v1.1 criteria.

#### **Duration of Response (DoR)**

DoR is defined as the time (in months) from date of first documented evidence of confirmed CR or PR to the date of first documented PD, as assessed by the investigator per RECIST v1.1 criteria, or to the date of death due to any cause among subjects with a BOR of confirmed CR or PR. Subjects who have not shown disease progression or died at the time of analysis will be considered censored as of the date of their last evaluable disease assessment. Censoring rules will follow those for PFS, specified in Table 3.

#### **Progression-Free Survival (PFS)**

PFS is defined as the time (in months) from the date of first dose until the date of first documented PD, as assessed by the investigator per RECIST v1.1 criteria, or date of death due to any cause, whichever occurs first. Subjects who have not shown disease progression or died at the time of analysis will be considered censored as of the date of

201973

their last evaluable disease assessment. Rules for determining the dates of PFS events and censoring are described in Table 3.

Table 3 – Assignments of Progression and Censoring Dates for PFS Analysis

| Scenario | Date of Event (PD<br>and/or Death) or<br>Censored | Event (PD<br>and/or Death)<br>or Censored |
|---|---|---|
| No adequate baseline assessments <sup>1</sup> and subject has not progressed or died (if the subject has progressed/died, follow the rules for death indicated at the bottom of the table). Note that PD may be documented in the RS (Response) or DS (Disposition) dataset. | First dose | Censored |
| No post-baseline assessments and subject has not died (if the subject has died, follow the rules for death indicated at the bottom of the table) and subject has no documented PD in DS dataset. | First dose | Censored |
| PD/death documented before any new anti-<br>cancer therapy is received. Note that this<br>includes PD/death at baseline or without<br>adequate assessments. | Date of assessment of PD <sup>2</sup> or date of death, whichever occurs first | Event |
| With post-baseline assessment(s) but no documented PD/death or new anti-cancer therapy. | Date of last 'adequate' assessment of response <sup>1</sup> | Censored |
| No adequate post-baseline assessment before start of new anti-cancer therapy and no PD documented in DS dataset. | First dose | Censored |
| With adequate post-baseline assessment(s) and new anti-cancer therapy started but without PD documented <sup>3</sup> | Date of last 'adequate'<br>assessment of response <sup>1</sup><br>(prior to starting new<br>anti-cancer therapy) | Censored |
| Death or PD documented in RS or DS dataset (without prior or new anti-cancer therapy) after two or more missed consecutive scheduled assessments | Date of last 'adequate'<br>assessment of response <sup>1</sup><br>(prior to missed<br>assessments) or date of<br>first dose without<br>'adequate' assessment <sup>1,4</sup> | Censored |

<sup>&</sup>lt;sup>1</sup> An adequate assessment is defined as a scheduled or unscheduled assessment in which the Investigator determines a disease response of CR, PR, or SD.

<sup>&</sup>lt;sup>2</sup> Equals the earliest of (a) date of radiological assessment showing new lesion (if progression is based on new lesion), or (b) date of radiological assessment showing unequivocal progression in non-target lesions,

201973

or (c) date of last radiological assessment of measured lesions (if progression is based on increase in sum of measured lesions).

<sup>3</sup> If documentation of PD and start of new anti-cancer therapy occur on the same day, PD will be assumed to have occurred first (i.e., prior to new therapy), with PD reported as the outcome and the assessment date reported as the event date.

<sup>4</sup> Relevant if the previous assessment is (a) earlier than Day 274 and the difference between PD/death and last adequate assessment is >126 days, or (b) between Day 274 and Day 344 and the difference between PD/death and last adequate assessment is >154 days, or (c) after Day 344 and the difference between PD/death and last adequate assessment is >182 days. Note that scheduled disease assessment window is +/-7 days.

### 7.2. Summary Measures

#### **Objective Response Rate (ORR)**

The number and percentage (representing ORR) of subjects in the population who show a BOR of confirmed CR or PR will be presented with exact 95% CI for ORR. Subjects with unknown or missing responses will be considered to be non-responders (i.e., subjects will be included in the denominator when calculating percentage). A spider plot of percent change from baseline in target lesions over time per subject and a waterfall plot of maximum percent reduction from baseline in tumour measurement per subject will be provided.

#### **Disease Control Rate (DCR)**

The number and percentage (representing DCR) of subjects in the population who show a BOR of confirmed CR, confirmed PR, or SD lasting ≥6 months will be presented with exact 95% CI for DCR. Subjects with unknown or missing responses will be treated as non-responders (i.e., subjects will be included in the denominator when calculating percentage).

#### **Duration of Response (DoR)**

Given a sufficient number of responses, DoR will be summarised using the Kaplan-Meier method. The median and 25<sup>th</sup> and 75<sup>th</sup> percentiles of DoR will also be estimated, with their corresponding 95% CIs estimated using the Brookmeyer-Crowley method (1982).

#### **Progression-Free Survival (PFS)**

PFS will be estimated using the Kaplan-Meier method. The median and 25<sup>th</sup> and 75<sup>th</sup> percentiles of PFS will also be estimated, with their corresponding 95% CIs estimated using the Brookmeyer-Crowley method (1982). A Kaplan Meier curve may also be produced, if the data warrant.

# 7.3. Population of Interest

Efficacy analyses will be based on the Modified All Treated Population, unless otherwise specified.

201973

### 7.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints/variables defined in Section 7.1 will be summarised using descriptive statistics, graphically presented (if appropriate), and listed.

| Primary Statistical Analyses | |
|---|---|
| Endpoint(s) | Method of Analysis |
| ORR | Percentage, Exact 95% CI |
| Secondary Statistical Analyses | |
| Endpoint(s) | Method of Analysis |
| DCR | Percentage, Exact 95% CI |
| DoR | Kaplan-Meier median and 25th and 75th percentiles,<br>Brookmeyer-Crowley 95% CIs (if data warrant) |
| PFS | Kaplan-Meier median and 25th and 75th percentiles,<br>Brookmeyer-Crowley 95% CIs (if data warrant) |

#### 8. SAFETY ANALYSES

Safety analyses will be based on the All Treated Population, unless otherwise specified. The results of all safety analyses will be presented by subject subgroup, defined by the combination of dose level, prior treatment, timing of a progressive disease response to prior treatment, and evidence of bone-only disease (see Section 5.5.2, Examination of Subgroups).

# 8.1. Adverse Events Analyses

Analyses of AEs, including summaries of all AEs, SAEs, and other significant AEs, will be based on GSK Core Data Standards. Moreover, all analyses will be performed on treatment-emergent AEs (TEAEs) only (see Section 15.4.3 for definition). The details of the planned displays are provided in Appendix 11: List of Data Displays.

All AEs will be coded by the Medical Dictionary for Regulatory Activities (MedDRA) System Organ Class (SOC) and Preferred Term (PT), as well as graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0.

Several summaries of AEs will be produced, including counts and percentages of subjects with:

- Any AE.
- Non-serious AEs.
- AEs related to study treatment (any, GSK525762, fulvestrant).
- AEs of Grade 3-4.

201973

- Grade 3-4 AEs related to study treatment (any, GSK525762, fulvestrant).
- AEs leading to permanent discontinuation of study treatment (any, GSK525762, fulvestrant).
- AE leading to dose reductions of study treatment (any, GSK525762, fulvestrant).
- AEs leading to dose interruptions/delays of study treatment (any, GSK525762, fulvestrant).
- SAEs.
- SAEs related to study treatment (any, GSK525762, fulvestrant).
- Non-fatal SAEs related to study treatment (any, GSK525762, fulvestrant).
- Dose-limiting toxicities.

A summary of common non-serious AEs (those that occur in ≥5% of subjects) will be provided (no rounding for the percentage will be used in terms of 5% threshold; e.g., events with 4.9% incidence rate will not be included in this table). This summary will contain the numbers and percentages of subjects per common non-serious adverse event. This summary table and those bulleted above will be displayed by SOC and PT.

A summary of the numbers and percentages of subjects with any AEs by maximum grade will be produced. At the subject level, a conservative approach will be taken to compute the maximum grade of AEs. Specifically, when grade is missing for one or more AEs for a single subject, the subject's maximum grade will be considered unknown. AEs will be sorted by MedDRA PT in descending order of total incidence. The summary will use the following algorithms for counting the subject:

- <u>PT row</u>: Subjects who experience multiple AEs of the same PT but with different grades will only be counted once with the maximum grade.
- Any event row: Each subject with at least one AE will be counted only once at the maximum grade no matter how many events they have.

In addition, the frequency and percentage of AEs (all grades) will be summarised and displayed in two ways: (1) in descending order of total incidence by MedDRA PT only and (2) in descending order of total incidence by MedDRA SOC x PT. In the SOC row, the number of subjects with multiple events of the same SOC will be counted only once.

Separate summaries will be provided for study treatment-related AEs, including GSK525762-related, fulvestrant-related, and any treatment-related (i.e., GSK525762 or fulvestrant-related) AEs. A study treatment-related AE is defined as an AE for which the investigator classifies the relationship to study treatment as "Yes". A worst-case scenario approach will be taken to handle missing relatedness data. That is, the summary table will include events with the relationship to study treatment as "Yes" or missing. The summary table will be displayed in descending order of total incidence by PT only. A summary of study treatment-related AEs by maximum grade will also be provided.

A summary of the number of subjects who experience DLTs will be provided. Lastly, all AEs, including DLTs, will be described in subject-level data listings.

201973

### 8.2. Adverse Events of Special Interest Analyses

A comprehensive list of MedDRA terms based on clinical review will be used to identify each type of AE of special interest (AESI). These AESIs are not defined in the protocol but are noted in the Investigational Brochure. Changes to the MedDRA dictionary may occur between the start of the study and time of reporting, and emerging data from ongoing studies may highlight additional AESIs. Therefore, the specific AESIs to be studied and the list of terms to be used per AESI will be based on Safety Review Team agreements that are in place at the time of database lock. Details of the planned displays are provided in Appendix 11: List of Data Displays.

AESIs will include, but may not be limited to, the following categories:

- Haematopoietic thrombocytopenia, Standardised MedDRA Query (SMQ)
- Haemorrhages [excluding laboratory terms] [NARROW] SMQ
- Anaemias nonhaemolytic and marrow depression, High Level Group Term (HLGT)
- Torsade de pointes/QT prolongation [NARROW] SMQ
- Drug related hepatic disorders comprehensive search [NARROW] SMQ
- Renal Preferred Terms

The PTs for AESIs will be provided by the GSK525762 Pharma Safety representative before DBR, based on the most up-to-date MedDRA version.

The number and percentage of subjects with AESIs will be summarised by AESI category, PT, and maximum toxicity grade in one table. A summary and a listing of event characteristics for each AESI category will also be provided, including number of subjects with any event, number of events, number of subjects with any serious event, number of subjects with any study treatment-related event, outcome of the event, maximum grade, and action taken for the event. The percentage of subjects with an AESI will be calculated using the total number of subjects as the denominator. The percentages of subjects associated with individual event characteristics will be calculated using the number of subjects with any AESI as the denominator. At a subject level, a worst-case approach will be applied for determining event outcome and maximum grade. That is, a subject with multiple AESIs will be counted only once based on the worst case from all AESIs experienced by the subject. For action taken to an event, subjects will be counted once per action. For example, if a subject has an event leading to both reduction of the study treatment dose and discontinuation of the study treatment, the subject will be counted once under both actions.

For each category of AESI, a summary of time to onset (in days) and duration of first occurrence (in days) will be provided, with each analysed as both a continuous and a categorical variable. Time to onset will be summarised within categories of 1-14 days, 15-28 days, and >28 days, and duration of first occurrence will be summarised within categories of 1-5 days, 6-10 days, and >10 days.

201973

#### 8.3. Deaths and Serious Adverse Events

For any subject who withdraws consent, no data after the date of consent withdrawal from this subject, including death, should appear in the database, which should be part of the data cleaning process.

All deaths will be summarised based on the number and percentage of subjects in the population. Within this summary, subjects will be classified by time of death relative to last dose of medication (>30 days vs. ≤30 days) and primary cause of death (disease under study, SAE related to study treatment, or other). A subject-level data listing will be generated to disclose the details of all death events.

All SAEs will be tabulated based on the number and percentage of subjects from the population who experience the specific SAE. Multiple summary tables will be generated, with statistics displayed in descending order of total incidence per PT only.

A study treatment-related SAE is defined as an SAE for which the investigator classifies the relationship to study treatment as "Yes". A worst-case scenario approach will be taken to handle missing relatedness data. That is, summary tables will include events with the relationship to study treatment as "Yes" or missing.

SAEs will be included in the listing of all AEs, and separate supportive listings with subject-level details will be generated for both fatal and non-fatal SAEs.

### 8.4. Adverse Events Leading to Discontinuation of Study Treatment and Other Significant Adverse Events

The following categories of AEs will be summarised separately in descending order of total incidence by PT only, and separate supportive listings will be generated with subject-level details for subjects with:

- AEs leading to permanent discontinuation of study treatment (any, GSK525762, or fulvestrant).
- AEs leading to dose interruptions/delays of study treatment (any, GSK525762, or fulvestrant).
- AEs leading to dose reductions of study treatment (any, GSK525762, or fulvestrant).

### 8.5. Extent of Exposure

Details of the extent of exposure to GSK525762 and fulvestrant will be both summarised and listed separately.

#### GSK525762:

The duration of exposure to study treatment in months (from first day of treatment to end of treatment in Phase I) will be summarised. Descriptive statistics, including mean, median, standard deviation, minimum, and maximum, will be computed for duration of study treatment. In addition, treatment duration will be summarised within the following categories: <3 months, 3 months to <6 months, 6 months to <12 months, and ≥12 months.

201973

The subject's average daily dose, defined as the cumulative dose divided by the duration of exposure for each subject, will be summarised.

Dose reductions will be summarised by number of reductions and number and percentage within categories of reason for reduction. Dose interruptions/delays will be summarised by number of interruptions/delays, reasons for interruption/delay, and duration of interruption/delay (in days). Descriptive statistics, including mean, standard deviation, median, minimum, and maximum, will be computed for interruption/delay duration, and the number and percentage of subjects within the interruption/delay duration categories of <7, 7-14, and >14 days will also be computed. A summary of dose escalation will also be provided, if applicable. All dose modifications (reductions, interruptions/delays, and escalations) will be listed separately.

#### **Fulvestrant:**

Duration of exposure, as well as cumulative dose and dose intensity (defined in Section 15.6.3), will be summarised for fulvestrant using descriptive statistics for a continuous variable.

Dose reductions will be summarised by number of reductions and number and percentage within categories of reason for reduction. Dose delays will be summarised by number of delays, number and percentage within categories of reason for delay, and duration of delay (in days). Descriptive statistics, including mean, standard deviation, median, minimum, and maximum, will be computed for delay duration. Missed doses will be summarised by number of missed doses and number and percentage within categories of reason for missed dose.

These summaries of dose modifications will be provided only if the data warrant. All dose reductions, interruptions/delays, and missed doses will be listed separately.

# 8.6. Pregnancies

Details of all pregnancies will be collected after the start of study treatment and until at least 90 days post-last dose of study drug. While pregnancy itself is not considered to be an AE or SAE, any pregnancy complication or elective termination of a pregnancy for medical reasons will be recorded as an AE or SAE. If a subject should become pregnant while on study, then information describing the pregnancy will be included in the narratives, and no separate table or listing will be produced.

# 8.7. Clinical Laboratory Analyses

Laboratory tests, including clinical chemistry, haematology, urinalysis, and liver function tests, will be based on GSK Core Data Standards. Details of the corresponding planned displays can be found in Appendix 11: List of Data Displays. Laboratory tests performed for the assessment of toxicity will include the following:

201973

Figure 2 – Clinical Laboratory Tests

| Clinical Chemistry |
|---|
| Sodium |
| Fasting Glucose |
| Potassium |
| Magnesium |
| Chloride |
| Calcium (total and ionized) |
| Total Carbon Dioxide |
| Total Protein |
| Blood Urea Nitrogen |
| Albumin |
| Creatinine |
| Hematology |
| White Blood cell count |
| Hemoglobin |
| Platelet count |
| Automated White Blood Cell Differential: |
| Neutrophils |
| Lymphocytes |
| Monocytes |
| Eosinophils |
| Basophils |
| Liver Function |
| Bilirubin (Total and, if Total is abnormal, then Direct needed) |
| Aspartate Aminotransferase (AST) |
| Alanine Aminotransferase (ALT) |
| Alkaline Phosphatase |
| Urinalysis |
| Specific gravity |
| рН |
| Glucose |
| Protein |
| Blood |
| Ketones |
| Microscopic examination (if urinalysis is abnormal) |
| Cardiac |
| Troponin (I or T), may be collected at central laboratory if local draw is not possible |
| N-terminal pro b-type natriuretic peptide (NT-proBNP) |
| Fasting Lipid Panel (Total Cholesterol, LDL, HDL, Triglycerides) |
| Other |
| Coagulation: |
| Prothrombin Time/Internal Normalized Ratio (INR) |
| Partial Thromboplastin Time (or Activated Partial Thromboplastin Time [aPTT]) |
| Fibrinogen |
| Factor VII Assay |
| Endocrine: |

201973

| Free Thyroxine 4 (Free T4) |
|--------------------------------------------------------|
| Hemoglobin A1c |
| FSH (for pre- and peri-menopausal subjects only) |
| Estradiol (for pre- and peri-menopausal subjects only) |
| Safety Screening: |
| HIV |
| HbSag |
| HCV antibody |
| Pancreatic Markers: |
| Amylase |
| Lipase |

A summary of laboratory values and derived change-from-baseline values by scheduled visit will be provided, using mean, median, standard deviation, minimum and maximum. Summaries of laboratory data will also be provided by maximum toxicity grade, using reported grades based on NCI-CTCAE v4.0. For any subject, a missing baseline grade will be assumed as grade 0.

Summaries of worst-case grade increase from baseline grade will be provided for all lab tests that are gradable by NCI-CTCAE v4.0. These summaries will display the number and percentage of subjects with a maximum post-baseline grade increasing from their baseline grade. Any increase in grade from baseline will be summarised along with any increase to a maximum grade of 3 and any increase to a maximum grade of 4.

Summaries will also include grade increase from baseline by scheduled visit. For laboratory tests that are graded for both low and high values, summaries will be generated separately and labeled by direction (e.g., low and high sodium level will be summarised as hyponatremia and hypernatremia, respectively).

For lab tests that are not gradable by NCI-CTCAE v4.0, summaries of worst-case changes from baseline with respect to normal range will be generated. Decreases to low, changes to normal or no changes from baseline, and increases to high will be summarised at each scheduled visit as well as for the worst-case post-baseline results. If a subject has a decrease to low and an increase to high during the same time interval, then the subject is counted in both the "Decrease to Low" categories and the "Increase to High" categories. In addition, the summary will include worst-case changes from baseline with respect to normal range by scheduled visits.

Separate summary tables for haematology, chemistry, liver function, urinalysis, and coagulation laboratory tests will be produced.

A supporting listing of laboratory data for subjects with abnormalities of potential clinical concern will be provided, as will a separate listing of laboratory data with character values.

Detailed derivation of baseline assessment is specified in Section 5.3, Baseline and Post-Baseline Definitions.

201973

Unless otherwise specified, the denominator used for computing percentages will be based on the number of subjects with non-missing values for the given scheduled visit.

Dipstick test results will be summarised at each scheduled visit. A supporting listing with subject level details will be provided.

Although all data will be reported according to the nominal visit for which they were recorded (i.e., no visit windows will be applied), summaries by visit will include data from scheduled assessments only. Unscheduled assessment data will be incorporated into "worse-case post-baseline" summaries, which capture the worst case across all scheduled and unscheduled visits following first dose of study treatment.

### 8.7.1. Analyses of Liver Function Tests

In addition to chemistry laboratory summaries and listings incorporating bilirubin (total and direct), aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase results, a summary and a listing of liver monitoring/stopping events defined by liver chemistry will be provided.

A summary and a listing of hepatobiliary laboratory abnormalities, including possible Hy's Law cases, will also be provided. Possible Hy's law cases will be defined as any event of either: (a) ALT  $\geq$ 3 × the upper limit of normal (ULN) and bilirubin  $\geq$ 2 × ULN (>35% direct bilirubin) or (b) ALT  $\geq$ 3 × ULN and INR >1.5, if INR is measured. Total bilirubin  $\geq$ 2 × ULN can be within 28 days following the ALT elevation and, if direct bilirubin is available on the same day, it must be  $\geq$ 35% of total bilirubin.

### 8.8. Other Safety Analyses

The analyses of non-laboratory safety test results, including those from vital signs, performance status, ECG, and ECHO/MUGA assessments, will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 11: List of Data Displays.

# 8.8.1. Vital Signs

Raw vital sign values, as well as computed changes from baseline, will be summarised by scheduled visit using mean, median, standard deviation, minimum and maximum.

In addition, vital sign values will be categorized as follows:

- Systolic blood pressure (BP; mmHg): Grade 0 (≤120), Grade 1 (>120 <140), Grade 2 (≥140 <160) and Grade 3 (≥160)
- <u>Diastolic BP (mmHg)</u>: Grade 0 (≤80), Grade 1 (>80 <90), Grade 2 (≥90 <100), and Grade 3 (≥100)
- Heart rate (beats/min): <60, 60-100, and >100
- Respiratory rate (breaths/min):  $<12, \ge 12 \le 18, >18 \le 25, \text{ and } >25$
- Temperature (°C):  $\leq 35, > 35 \leq 38, \geq 38$
201973

Summaries of increase in vital signs from the baseline with respect to the categories defined above will be performed. These summaries will display the number and percentage of subjects in the population with any grade increase, an increase to grade 2, and an increase to grade 3 at each scheduled visit and at the visit showing the worst-case post-baseline results.

#### 8.8.2. Performance Status

Eastern Cooperative Oncology Group (ECOG) performance status will be summarised at baseline and each post-baseline scheduled visit. Summaries will include the numbers and percentages of subjects in the population at each planned assessment time. A summary of change-from-baseline by scheduled visit will be generated, as will a summary of the worst-case and best-case post-baseline changes during the study (i.e., using categories of improved, no change, and deteriorated). A supporting listing will also be provided.

#### 8.8.3. ECG

Per protocol, triplicate 12-lead ECGs will be obtained, prior to dosing, during the study using a standard 12-lead ECG machine that automatically calculates heart rate and measures PR, QRS, QT and QTcF intervals. The baseline QTcF value will be computed as the mean of the triplicate Week 1 Day 1 pre-dose QTcF results (see Section 5.3, Baseline and Post-Baseline Definitions). If these results are not available, then the mean QTcF of the screening triplicate ECG results will be used.

A summary of the number and percentage of subjects with normal, abnormal clinically significant, and abnormal not clinically significant ECG findings will be displayed by scheduled visit, as well as for the worst-case post-baseline assessment.

Change from baseline in ECG values will be summarized at each scheduled assessment time and for the worst-case post-baseline. Only the post-baseline assessments that used the same source (i.e., local or central cardiologist read) as the baseline assessments will be used to derive the change from baseline; data from two sources will not be combined.

QTcF prolongation will be monitored throughout the study. QTcF values will be rounded to the integer and categorized into the following ranges: Grade 0 (<450 msec), Grade 1 (450-480 msec), Grade 2 (481-500 msec), and Grade 3 (≥501 msec).

Summaries of grade increase will be provided. These summaries will display the number and percentage of subjects in the population with any grade increase, an increase to grade 2, and an increase to grade 3 at each scheduled visit and at the visit showing the worst-case post-baseline results. Missing baseline grade will be assumed as grade 0.

Changes in QTc values will be categorized into ranges of clinical concern, namely differences of 31-60 msec and >60 msec from baseline. A summary of change in QTc value will display the number and percentage of subjects in each range of clinical concern per scheduled visit and at the visit showing the worst-case post-baseline results. Subjects with missing baseline values will be excluded from this summary.

Listings of all ECG results and all abnormal ECG findings will be provided.

201973

#### 8.8.4. LVEF

Both absolute and relative change from baseline in LVEF will be summarised at each scheduled visit and at the visit showing the worst-case post-baseline results. Only the post-baseline assessments that used the same method (ECHO or MUGA) and source (local or central) as the baseline assessments will be used to derive the change from baseline. Absolute change from baseline will be categorized as follows:

- No change or any increase (i.e., increases of 0 to <10%, 10 to <20%, and  $\ge 20\%$ )
- Any decrease (i.e., decreases of >0 to <10%, 10 to <20%, and  $\ge 20\%$ )
- Decrease  $\geq 10\%$  and  $\geq$  lower limit of normal (LLN)
- Decrease >10% and < LLN
- Decrease  $\geq 20\%$  and  $\geq LLN$
- Decrease >20% and < LLN

Relative change from baseline will be categorized as follows:

- Decrease  $\geq 20\%$  and  $\geq LLN$
- Decrease ≥20% and < LLN

A listing of all LVEF results will be produced, including both absolute and relative changes from baseline.

#### 8.8.5. Liver Events

For any liver events that occur during the study, the Roussel Uclaf Causality Assessment Method (RUCAM) score will be derived and incorporated into a listing of data describing liver monitoring/stopping events. The score incorporates whether the subject was age 55 years or older, the subject became pregnant, liver imaging was normal or not, a biopsy was taken or not, fasting or significant dietary change occurred, and the subject took any unconventional medications, as well as the relative timing of the event (i.e., while on treatment vs. after stopping treatment) and computed durations from first dose to start of the liver event.

#### 9. PHARMACOKINETIC ANALYSES

# 9.1. Primary Pharmacokinetic Analyses

### 9.1.1. Endpoint / Variables

# 9.1.1.1. Drug Concentration Measures

Two major metabolites of GSK525762, GSK3529246 and GSK3536835, have been observed in humans. GSK3536835 was found to be unstable under bioanalytical conditions. Therefore, the two major active metabolites were measured together following full conversion of GSK3536835 to GSK3529246 prior to analysis and the active metabolites (GSK3529246 + GSK3536835) are reported as one entity, GSK3529246.

201973

Concentrations of GSK525762, active metabolites (GSK3529246), and GSK525762 total active moiety (i.e. GSK525762 + GSK3529246 after conversion from ng/mL to nM concentrations) and fulvestrant will be listed for each subject.

Summaries of plasma concentration will be produced separately for GSK525762 in both ng/mL and nM, active metabolites (GSK3529246) in both ng/mL and nM and the total active moiety of GSK525762 (GSK525762 + GSK3529246 after conversion to nM concentrations) in nM. Plasma concentration-time data will be summarized using descriptive statistics (n, mean, SD, median, minimum and maximum) by planned relative assessment time.

Mean/median plots of concentration (GSK525762 in nM, GSK3529246 in nM, and total active moiety in nM on the same plot) over time will be provided for each analyte using actual elapsed time for Week 1 and Week 3 for GSK525762, GSK3529246, and Total active moiety and using overall duration of the study for fulvestrant.

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 13.5.3, Reporting Standards for Pharmacokinetic) for details of displays.

#### 9.1.1.2. Derived Pharmacokinetic Parameters

The PK parameters presented in the table below will be derived during programming. This will be the responsibility of the Statistics and Programming group at PAREXEL under the direction of the Clinical Pharmacology Modeling and Simulation (CPMS) Department at GSK.

The parameters will be determined from the concentration-time data for GSK525762 (in ng/mL), active metabolites (GSK3529246 in ng/mL), and total active moiety (i.e. GSK525762 + GSK3529246 in nM), as data permits.

The molecular weight of GSK525762 is 424 g/mol, and the molecular weight of GSK3529246 is 396 g/mol. The total active moiety concentration in nmol/L will be computed as (GSK525762 concentration in ng/mL / molecular weight of 424 x 1000) + (GSK3529246 concentration in ng/mL / molecular weight of 396 x 1000).

| Parameter | Parameter Description |
|---|---|
| C <sub>max</sub> | Maximum observed concentration; determined directly from the concentration-time curve. |
| T <sub>max</sub> | Time from first administration to occurrence of $C_{\text{max}}$ ; determined directly from the concentration-time curve. |
| Ст | Also referred to as "C <sub>trough</sub> "; observed concentration at the end of a dosing interval, immediately before the next administration; determined directly from the concentration-time curve. |

**NOTE:** Additional parameters may be included as required

201973

#### 9.1.2. Summary Measure

Summaries of plasma concentration will be produced separately for GSK525762 in both ng/mL and nM, active metabolites (GSK3529246) in both ng/mL and nM and the total active moiety of GSK525762 (GSK525762 + GSK3529246 after conversion to nM concentrations) in nM, and fulvestrant.

Plasma concentration-time data will be summarised using descriptive statistics (n, mean, SD, median, minimum and maximum) by planned relative assessment time. Mean and/or median values will be plotted over time using nominal/scheduled visit.

Concentration-time profiles for GSK525762, GSK3529246, and the total active moiety of GSK525762 will be overlaid on the same plot conversion to nM concentrations.

The PK parameters described in Section 9.1.1.2 will also be summarised descriptively (using mean, SD, median, minimum, maximum, geometric mean with SD, coefficient of variation [CV], and 95% CI of log-transformed parameters, if applicable), separately for GSK525762, active metabolites (GSK3529246), and the total active moiety of GSK525762.

# 9.1.3. Population of Interest

The primary PK analyses will be based on the PK Population, unless otherwise specified.

#### 10. PHARMACODYNAMIC ANALYSIS

The pharmacodynamic analyses will be detailed in a Pharmacodynamic RAP supplement and will not be discussed as part of this RAP.

#### 11. OTHER STATISTICAL ANALYSES

#### 11.1. Value Evidence and Outcomes

The value evidence and outcomes analyses will be based on the Modified All Treated Population, unless otherwise specified. All summaries and data listings will use treatment labels as specified in Section 5.1, Study Treatment and Sub-group Display Descriptors.

Summaries of raw values and absolute change-from-baseline values from the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC-QLQ-C30) and Breast-23 (EORTC-QLQ-BR23) scales will be provided in tables. Summaries of raw values and absolute change-from-baseline values from Patient Reported Outcomes Common Terminology Criteria for Adverse Events (PRO-CTCAE) will be provided in tables. Single items from EORTC-QLQ-C30, EORTC-QLQ-BR23, and PRO-CTCAE will be provided in listings.

Baseline will be defined as the visit prior to the start of Week 1 Day 1 dosing. Details of data displays are presented in Appendix 11: List of Data Displays.

201973

# 12. REFERENCES

Brookmeyer R, Crowley J. A confidence interval for the median survival time. Biometrics, 1982; 38:29-41.

Aaronson, N. K., Ahmedzai, S., Bergman, B., Bullinger, M., Cull, A., Duez, N. J., Takeda, F. (1993). The European Organization for Research and Treatment of Cancer QLQ-C30: A Quality-of-Life Instrument for Use in International Clinical Trials in Oncology. *JNCI: Journal of the National Cancer Institute*, 85(5), 365-376.

201973

# 13. APPENDICES

# 13.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

Protocol deviations will be tracked by the study team throughout the study in accordance with the Protocol Deviation Specification document.

# 13.1.1. Exclusions from Per Protocol Population

No Per Protocol Population will be defined or used for this study.

# 13.2. Appendix 2: Schedule of Activities

Refer to Protocol Section 7, Study Assessments and Procedures.

# 13.3. Appendix 3: Assessment Windows

No assessment windowing will be applied in this study.

# 13.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

# 13.4.1. Study Phases

Disease assessments and AEs, SAEs, death, laboratory data, vital signs, ECGs, ECHO/MUGA scans, ECOG results, and other safety domains will be assigned to the treatment phases defined below. Partial dates will be imputed into full dates, if applicable, for slotting data to the appropriate categories below. Flag variables (time in relation to study treatment) indicating the study time periods will be added to these datasets.

Assessments and events will be classified according to the time of occurrence relative to Study Treatment Start Date.

| Treatment<br>Phase | Definition |
|---|---|
| Pre-Treatment | Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ Date ≤ Study Treatment Stop Date |
| Onset Time<br>Since 1 <sup>st</sup> Dose<br>(Days) | <ul> <li>If Treatment Start Date &gt; AE Onset Date = AE Onset Date - Treatment Start Date</li> <li>If Treatment Start Date ≤ AE Onset Date = AE Onset Date - Treatment Start Date +1</li> <li>Missing otherwise.</li> </ul> |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |

**NOTES:** If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.

#### 13.4.2. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment.

### 13.4.2.1. Treatment States for Disease Response Data

| Treatment<br>State | Definition |
|---|---|
| Time to | (Date of Progression or Date of Last Disease Assessment) – Study |
| Progression | Treatment Start Date + 1 |
| Time to | (Date of First Partial or Complete Response of a Confirmed Partial or |
| Response | Complete Response) – Study Treatment Start Date + 1 |
| Duration of | (Date of Progression or Date of Death) – (Date of First Partial or Complete |
| Response | Response of a Confirmed Partial or Complete Response) + 1 |

201973

# 13.4.3. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | If AE onset date is on or after treatment start date and on or before 30 days after treatment end date. |
| | • Study Treatment Start Date ≤ AE Start Date ≤ (Study Treatment End Date + 30 days). |
| | If AE onset date is prior to treatment start date and toxicity grade changes to worsening on or after treatment start date and on or before treatment end date + 30 days. |
| | • AE onset Date < Study Treatment Start date and Study Treatment Start Date ≤ AE Worsening Date ≤ (Study Treatment End Date + 30 days). |
| Drug-Related | If relationship is marked 'YES' on Inform/CRF (or if value is missing). |

#### **NOTES:**

- If completely missing start dates, then the AE will be considered as TEAE.
- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

201973

# 13.5. Appendix 5: Data Display Standards & Handling Conventions

# 13.5.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | US1SALX00259 |
| HARP Compound | GSK525762\mid201973 |
| <b>Analysis Datasets</b> | |
| Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 & ADaM IG Version 1.1). | |
| Generation of RTF Files | |
| RTF files will be generated for SAC and IA upon request. | |

# 13.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:
  - https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - o 4.03 to 4.23: General Principles
  - o 5.01 to 5.08: Principles Related to Data Listings
  - o 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report.
   All subject level listings should be located in the modular appendices as ICH or non-ICH listings

#### Formats

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DPs) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DPs.

#### **Planned and Actual Time**

• Reporting for tables, figures and formal statistical analyses:

201973

- o Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
- The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - o Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables, except in cases where worst-case post-baseline is calculated.
- Unscheduled visits will not be included in figures, unless otherwise specified.
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| | • |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |
| · | |

# 13.5.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic C | Pharmacokinetic Concentration Data |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non-compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to SOP_00000314000: Non-compartmental Analysis of Clinical Pharmacokinetic Data. Note: Concentration values will be imputed as per GUI_51487. |
| ADPC data file | To create ADPC the SDTM PC domain dataset will be merged with the Subject-Level Analysis Dataset (to get demographic information) and with SDTM EX domain (to get reference timepoint date). Reference timepoint date will be populated for both study drug and active metabolite based on study treatment information from SDTM EX domain. To populate analysis values in ADPC (AVAL(C)) adjustments to the PCSTRESN will be done based on imputation rules from "Non-Compartmental Analysis of Pharmacokinetic Data, CPMS Global" document. |

201973

| | Total Moiety parameter will be added, along with concentrations of study drug and active metabolite, and derived as the sum of study drug and active metabolite concentrations converted to nM units. |
|---|---|
| | The molecular weight of GSK525762 is 424 g/mol and the molecular weight of GSK3529246 is 396 g/mol. The total active moiety concentration in nmol/L will be computed as (GSK525762 concentration in ng/mL / molecular weight of 424 x 1000) + (GSK3529246 concentration in ng/mL / molecular weight of 396 x 1000). |
| Descriptive | Refer to IDSL PK Display Standards. |
| Summary Statistics, Graphical Displays | Refer to IDSL Statistical Principle 6.06.1. |
| and Listings | <b>Note:</b> Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarised graphical displays only. Assign zero to NQ values. |
| Pharmacokinetic Pa | arameter Derivation |
| PK Parameters to<br>be Derived by PK<br>Programmer | The following PK parameters will be derived by the PK Programmer: $C_{max}$ , $T_{max}$ , and $C_{\tau}$ . |
| Pharmacokinetic Parameter Data | |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | Yes. Refer to Standards for Handling NQ Impacted PK Parameters. |

201973

## 13.6. Appendix 6: Derived and Transformed Data

#### 13.6.1. **General**

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but, if listed, all data will be presented.
- If multiple assessments on different days are reported for the same scheduled assessment, then the worst-case assessment for that scheduled assessment will be analysed.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from Study Treatment Start Date to Reference Date:
  - If Ref Date = Missing, then Study Day = Missing.
  - If Ref Date < Study Treatment Start Date, then Study Day = Ref Date Study Treatment Start Date.
  - o If Ref Data ≥ Study Treatment Start Date, then Study Day = Ref Date (Study Treatment Start Date) + 1.

#### **Change from Baseline**

- Absolute Change from Baseline = Post-Baseline Visit Value Baseline Value.
- Percent (i.e., Relative) Change from Baseline = ([Post-Baseline Visit Value Baseline Value] ÷ Baseline Value) x 100.

If either the Baseline or Post-Baseline Visit Value is missing, then both Absolute and Relative Change from Baseline are set to missing.

## **Date of Response**

For post-baseline disease assessments, the date of response (PR or better) is assigned to the earliest date of disease assessments showing the response (not to the date on which confirmation ultimately occurs); for other response categories not requiring confirmation (SD [or Non-CR/Non-PD], NE, PD), the date of response is also assigned to the earliest date of disease assessments showing the response.

#### **Date of New Anti-Cancer Therapy**

Derived as the earliest date of new anti-cancer therapy, radiotherapy (where applicable) or cancer-related surgical procedure (where applicable). Missing or partial dates will be imputed for derivation of new anti-cancer therapy following rules specified in Section 13.7.3.

201973

### 13.6.2. Study Population

#### Demographics

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - o Any subject with a missing day will have this imputed as day '15'.
  - o Any subject with a missing date and month will have this imputed as '30th June'.
  - o Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)]<sup>2</sup>

# **13.6.3.** Efficacy

#### **Primary Endpoint**

#### **Objective Response Rate (ORR)**

- Defined as the percentage of subjects in the population who demonstrate a Best Overall Response (BOR) of confirmed Complete Response (CR) or Partial Response (PR), as assessed by the investigator per RECIST v1.1 criteria.
- Subjects with unknown or missing response will be treated as non-responders (i.e., these subjects will be included in the denominator when calculating the percentage).

#### **Secondary Endpoints**

#### **Disease Control Rate (DCR)**

- Defined as the percentage of subjects in the population with a confirmed CR, confirmed PR, or Stable Disease (SD) lasting ≥6 months, as assessed by the investigator per RECIST v1.1 criteria.
- Subjects with unknown or missing response will be treated as non-responders (i.e., these subjects will be included in the denominator when calculating the percentage).

#### **Duration of Response (DoR)**

- Defined as the time (in months) from date of first documented evidence of confirmed CR or PR to the date of first documented progressive disease (PD), as assessed by the investigator per RECIST v1.1 criteria, or to the date of death due to any cause (whichever occurs first) among subjects with a BOR of confirmed CR or PR.
- Subjects who have not shown disease progression or died at the time of analysis will be considered censored as of the date of their last evaluable disease assessment, but censoring rules for other unique scenarios (e.g., receipt of new anti-cancer therapy) will adhere those rules defined for PFS.

#### **Progression Free Survival (PFS)**

- Defined as the time (in months) from the date of first dose until the date of first documented PD, as assessed by the investigator per RECIST v1.1 criteria, or date of death due to any cause, whichever occurs first.
- Subjects who have not shown disease progression or died at the time of analysis will be considered censored as of the date of their last evaluable disease assessment. Rules for determining the dates of PFS events and censoring are described in **Table 3**.

201973

# 13.6.4. Safety

#### **Adverse Events**

#### **AEs of Special Interest**

- Haematopoietic thrombocytopenia Standardised MedDRA Query (SMQ)
- Haemorrhages [excluding laboratory terms] [NARROW] SMQ
- Anaemias nonhaemolytic and marrow depression High Level Group Term (HLGT)
- Torsade de pointes/QT prolongation [NARROW] SMQ
- Drug related hepatic disorders comprehensive search [NARROW] SMQ
- Renal Preferred Terms

#### ECHO/MUGA

Only the post-baseline assessments that use the same method (i.e., ECHO or MUGA) and source (i.e., local or central read) as the baseline assessments will be used to derive the change from baseline. Data from different methods and sources should not be combined.

201973

#### **Extent of Exposure**

- Number of days of exposure to GSK525762 will be calculated based on the formula:
  - Duration of Exposure in Days = Treatment Stop Date Treatment Start Date + 1.
- Number of days of exposure to fulvestrant will be calculated based on the formulas:
  - Duration of Exposure in Days = ([Treatment Stop Date + 13] Treatment Start Date) +
     1, if the last dose date is the first two doses.
  - Duration of Exposure in Days = ([Treatment Stop Date + 27] Treatment Start Date) +
     1, if the last dose date is not the first two doses.
- Subjects who were not screen failures but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose for GSK525762 will be calculated based on the formula:
  - Cumulative Dose = Sum of (Number of Days x Total Daily Dose)
- The cumulative dose for fulvestrant will be calculated based on the formula:
  - Cumulative Dose = Sum of (Total Daily Dose)
- The relative dose intensity for GSK525762 will be calculated based on the formula:
  - $\circ$  Relative Dose Intensity (%) = (Dose Intensity / Planned Dose Intensity) x 100.

#### **Laboratory Parameters**

If a laboratory value that is expected to have a numeric value for summary purposes has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.

Example 1: 2 Significant Digits = '< x' becomes x -0.01

Example 2: 1 Significant Digit = '> x' becomes x + 0.1

Example 3: 0 Significant Digits = '< x' becomes x – 1

#### 13.6.5. Value Evidence and Outcomes

#### EORTC QLQ-C30 and EORTC QLQ-BR23

- Both the QLQ-C30 and the QLQ-BR23 are composed of multi-item scales and single-item
  measures. The QLQ-C30 includes a global health status/QoL scale, five functional scales,
  and nine symptom scales/items. The QLQ-BR23 includes five functional scales and four
  symptom scales/items.
- Each of the multi-item scales includes a different set of items; no item occurs in more than one scale.
- All the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
  - o Thus, a high score for the global health status/QoL represents a high QoL, and
  - o a high score for a functional scale represents a high/healthy level of functioning, but
  - o a **high score for a symptom scale/item** represents a *high level of symptomatology/problems*.
- The principle for scoring these scales is the same in all cases:
  - Estimate the average of the items that contribute to the scale to calculate the *raw score*.
  - Use a linear transformation to standardise the raw score, so that scores range from 0 to 100. A higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.

#### **Technical Summary**

In practical terms, if items  $I_1, I_2, ... I_n$  are included in a scale, the procedure is as follows:

(1) Calculate the raw score:



- (2) Apply the linear transformation to 0-100 to obtain the score *S*:
  - Global health status / QoL:
  - Functional scales:
  - Symptom scales / items:

Range is the difference between the maximum possible value of RS and the minimum possible value. Both questionnaires have been designed so that all items in any scale take the same range of values. Therefore, the range of RS equals the range of the item values. Most items are scored 1 to 4, giving range = 3. The exceptions are the QLQ-C30 items contributing to global health status/QoL, which are 7-point questions with range = 6, and the initial yes/no items on the earlier versions of the QLQ-C30 which have range = 1.

#### EORTC QLQ-C30

201973

| EORTC QLQ-C30 and EORTC QLQ-BR23 | | | | | |
|---|---|---|---|---|---|
| | Scale | Number of Items | Item<br>Range | Item<br>Numbers | Functional<br>Scales |
| CCI - This section contained Clinical C<br>which are protected by third party cop | Outcome Asses<br>yright laws and | sment data col | lection question | naires or indices | , |
| "Item range" is the difference | e between th | ne possible n | naximum and | d the minimu | m response to |
| individual items; most items | | | | | 1 |
| *Items for the scales marked | * are score | d positively | (i.e. "very m | uch" is best) | and therefore |
| use the same algebraic equation | on as for sy | mptom scale | | | |
| the algebraic equation for fun | ictioning sca | ues. | | | |
| | | ble if item | | .,, | |
| is i | not applicab | le if item 🛗 | s ' <mark>CCl</mark> | , | |
| EORTC QLQ-BR23 | T = - | T | 1 _ | 1 _ | |
| | Scale | Number of Items | Item<br>Range | Item<br>Numbers | Functional Scales |
| CCI - This section contained Clinical which are protected by third party cop | Outcome Asse | ssment data co | llection question | naires or indices | S, |
| - | | | | | |
| - | | | | | |
| _ | | | | | |
| - | | | | | |
| - | | | | | |
| - | | | | | |
| "Item range" is the difference | between th | e possible m | aximum and | the minimum | n response to |
| individual itams: most itams | | | | | 1 |

201973



#### **PRO-CTCAE**

- The response frequency distribution and proportion of subjects for each PRO-CTCAE item will be presented by visit. This should be grouped first by visit, then by related term.
- Subjects who do not have a response due to skipping patterns should be reported as "Not applicable". Other subjects who do not provide a response or have withdrawn from the study should be treated as missing data. The number of subjects who provide a response should be reflected in the number of observations for the sample.
- In addition to reporting the number and percent of subjects who have selected each response category, assign a value (see coding table below:

  CCI for CCI and calculate the mean (SD) and median values for all subjects who have a valid response for a given visit. Subjects with missing or incomplete data (either due to dropouts, or subjects who have not provided a response either due to missing data or skip patterns) should be excluded from calculating the mean and median.



- PRO-CTCAE responses should also be summarised by changes in health state. For each subject, compare their current response with the response from their prior assessment and determine whether their symptoms improved, worsened or were stable, based on the following criteria:
  - Improved = current response level < prior response level</li>
  - Worsened = current response level > prior response level
  - Stable = current response level = prior response level
- Due to conditional branching and skip patterns it is possible that a response option may be missing. In these cases, the lowest level would be imputed in order to calculate the state change. Subjects who have data missing for other reasons (missing data, drop out) will be excluded for any item/visit where they have missing data.
- In addition to reporting the response frequencies by visit, as suggested by the FDA, report the results of PRO-CTCAE alongside the corresponding clinician-graded CTCAE results.

201973

# PRO-CTCAE

- Categorize the highest level reported as either "Any Level" (subjects who had either a CTCAE or PRO-CTCAE response >0) or "High Level" (subjects who experienced ≥3 grade CTCAE or PRO-CTCAE response).
- Listings should include response values (0-4, null for missing) for all PRO-CTCAE Items by subject and visit.

# 13.7. Appendix 7: Reporting Standards for Missing Data

# 13.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>The study will be considered completed for purposes of final analysis when approximately 70% of enrolled subjects have died. However, as originally planned, the study can be stopped due to toxicity or futility before this time-point when there is enough evidence to conclude as such.</li> <li>Given current study status, the totality of Phase I data assessed at the interim analysis does not support continuing investigation of GSK525762 (molibresib) in combination with fulvestrant for the treatment of HR+/HER2- advanced or metastatic breast cancer patients. As interim data failed to demonstrate meaningful clinical benefit in this patient population, enrolment into the study is now closed and the study will not incorporate Phase II.</li> <li>With the implementation of Amendment 06, specific assessments and collection of survival follow-up data will no longer be required. The study will conclude when the last subject has completed/discontinued study treatment and completed the end of treatment visit.</li> <li>All available data from subjects who have withdrawn from the study will be listed, and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 13.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occur when any requested data are not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data are excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> |
| Responder<br>Analysis | • For endpoints which determine the percentage of responders, subjects with unknown or missing response will be treated as non-responders and will be included in the denominator when calculating the percentages. |

# 13.7.3. Handling of Missing and Partial Dates

Imputed partial dates can be used to derive study day, duration (e.g. duration of adverse events), or elapsed time variables. Imputed dates will not be used for deriving the last contact date in the overall survival analysis dataset.

201973

With the exception of new anti-cancer start date on the Oncology time to event analysis dataset and exposure end date on the Exposure analysis dataset, imputed dates will also not be stored on datasets.

Imputed dates will not be displayed in listings. However, where necessary, display macros may impute dates as temporary variables for the purpose of sorting data in listings only. In addition, partial dates may be imputed for 'slotting' data to study time periods or for specific analysis purposes as outlined below.

The partial date imputation will follow ADaM conventions. The ADaM approach is to populate the numeric date variables with the imputed date and add a flag variable to the dataset that indicates the level of imputation.

The flag variable can contain the values: blank, 'D', 'M', 'Y'.

blank: indicates that no imputation was done

D='Day': indicates that the day portion of the date is imputed

M='Month': indicates that the month and day portions of the date are imputed

Y='Year': indicates that the entire date (year, month, and day) is imputed

#### Example of date variables:

XYZD - character date variable

XYZDT - numeric date variable

XYZDTFL - flag variable

Details on imputing partial dates for specific datasets are outlined below.

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse Events | • The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: |
| | <ul> <li>Missing Start Day: First of the month will be used unless this is<br/>before the start date of study treatment; in this case the study<br/>treatment start date will be used and hence the event is considered<br/>On-treatment as per Appendix 4: Study Phases and Treatment<br/>Emergent Adverse Events.</li> </ul> |
| | <ul> <li>Missing Stop Day: Last day of the month will be used, unless this is<br/>after the stop date of study treatment; in this case the study<br/>treatment stop date will be used.</li> </ul> |
| | Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such |

201973

| Element | Reporting Detail |
|---|---|
| | events will be missing. If completely missing start dates, TEAE flag is Yes. |
| | Start or end dates of which are completely missing (i.e., no year specified) will remain missing, with no imputation applied. |
| Anti-Cancer<br>Therapy<br>(including<br>Radiotherapy)<br>and Surgical<br>Procedures | <ul> <li>Completely missing start dates will remain missing, with no imputation applied.</li> <li>Partial start dates will be imputed using the following convention: <ul> <li>If both month and day are missing, no imputation will be applied.</li> <li>If only day is missing: <ul> <li>If the month of partial date is the same as the month of last dosing date, minimum of (last dosing date + 1, last day of the month) will be used for the day.</li> <li>If the month of partial date is the same as the month of last disease assessment and the last disease assessment is PD, minimum of (last date of disease assessment + 1, last day of the month) will be used for the day.</li></ul></li></ul></li></ul> |
| Concomitant | <ul> <li>imputation applied.</li> <li>Partial dates for any concomitant medications recorded in the eCRF will</li> </ul> |
| Medications,<br>Medical<br>History, and<br>Blood Products | <ul> <li>be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> <li>The recorded partial date will be displayed in listings.</li> <li>No Imputation for completely missing start or end dates.</li> </ul> |
| Time to Event<br>and Response<br>for Anti-Cancer<br>Therapy, and,<br>where<br>applicable,<br>Radiotherapy<br>and Surgical<br>Procedures | <ul> <li>Start dates for subsequent anti-cancer therapy, radiotherapy (where applicable), and surgical procedures (where applicable) will be temporarily imputed in order to define event and censoring rules for progression-free survival, response rate, or duration of response (i.e. start date for new anti-cancer therapy). Dates will only be imputed when a month and year are available, but the day is missing. The imputed dates will not be stored on the anti-cancer therapy, radiotherapy, or surgical procedure datasets. The following rules will be used to impute the date when partial start dates are present on anti-cancer therapy radiotherapy, and/or surgical procedures datasets.</li> <li>No Imputation for completely missing start dates.</li> </ul> |

201973

| Element | Reporting Detail |
|---|---|
| | No imputation for missing start day and month (note: the eCRF should only allow for missing day). |
| | • If partial start date falls in the same month as the last dose of study treatment, then assign to earlier of (date of last dose of study treatment+1, last day of month). |
| | • If partial start date falls in the same month as the subject's last assessment and the subject's last assessment is progressive disease (PD), then assign to earlier of (date of PD+1, last day of month). |
| | • If both rules above apply, then assign to latest of the 2 dates. |
| | Otherwise, impute missing day to the first of the month. |
| | No imputation for partial end dates will be performed. |
| Exposure End Dates for | If treatment discontinuation date is missing, then assign exposure end date as the earliest of: |
| Subjects Who<br>Are Still on<br>Study at the | o date of the data cutoff, |
| | o date of withdrawal from the study, or |
| Time of Analysis | o death date. |
| 7 mary 515 | The imputed exposure end date will be used to calculate cumulative dose and exposure duration. |
| | The imputed exposure end date will be stored in the exposure analysis dataset and an exposure end date imputation flag variable will be derived indicating which exposure end date records are imputed. |
| | Imputed exposure end dates will also be stored on the study treatment end date variable. |
| | • For subjects who are still on study treatment, the on-therapy indicator variables (time in relation to study treatment) are assigned to on-therapy for all records where the 'dataset'.'date' is after or on the study treatment start date. |

#### 13.8. Appendix 8: Values of Potential Clinical Importance

#### 13.8.1. Laboratory Values

Reference ranges for all laboratory parameters collected throughout the study are provided by the laboratory. A laboratory value that is outside the reference range is considered either high abnormal (value above the upper limit of the reference range) or low abnormal (value below the lower limit of the reference range). Note: a high abnormal or low abnormal laboratory value is not necessarily of clinical concern. The laboratory reference ranges will be provided on the listings of laboratory data. Clinical laboratory test results outside of the reference range will be flagged in the listings.

To identify laboratory values of potential clinical importance, National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v4.0) will be used to assign grades to the relevant laboratory parameters. NCI-CTCAE v4.0 can be found at <a href="http://ctep.cancer.gov/reporting/ctc.html">http://ctep.cancer.gov/reporting/ctc.html</a>.

For laboratory data which are not listed in the NCI CTCAE v4.0, a summary of values outside the normal range will be provided.

13.8.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|-----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| | msec | ≥ 450 | < 481 |
| Absolute QTcF Interval | | ≥ 481 | < 501 |
| | | ≥ 501 | |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | <75 | >110 |
| Change from Baseline | | | |
| Decrease from Baseline QTcF | msec | > 30 | ≤ 60 |
| Decrease from Baseline QTCF | | > 60 | |
| Increase from Descline OTeE | msec | > 30 | ≤ 60 |
| Increase from Baseline QTcF | | > 60 | |

## 13.8.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| (Absolute) | | Lower | Upper |
| | | > 120 | < 140 (Grade 1) |
| Systolic Blood Pressure | mmHg | ≥ 140 | < 160 (Grade 2) |
| | | | ≥ 160 (Grade 3) |
| | mmHg | > 80 | < 90 (Grade 1) |
| Diastolic Blood Pressure | | ≥ 90 | < 100 (Grade 2) |
| | | | ≥ 100 (Grade 3) |
| Heart Rate | bpm | < 60 | > 100 |
| Temperature | Degrees C | ≤ 35 | ≥ 38 |

201973

# 13.8.4. Left Ventricular Ejection Fraction

| LVEF | Units | Clinical Concern Range |
|-------------------------------|-------|-----------------------------------|
| | | Increase $\geq 0$ and $< 10$ |
| | | Increase $\geq 10$ and $\leq 20$ |
| | % | Increase $\geq 20$ |
| | | Decrease > 0 and < 10 |
| Absolute Change from Deceline | | Decrease $\geq 10$ and $\leq 20$ |
| Absolute Change from Baseline | | Decrease ≥ 20 |
| | | Decrease $\geq 10$ and $\geq LLN$ |
| | | Decrease $\geq 10$ and $\leq LLN$ |
| | | Decrease $\geq 20$ and $\geq LLN$ |
| | | Decrease $\geq 20$ and $\leq LLN$ |
| Palativa Changa from Pagalina | | Decrease $\geq 20$ and $\geq LLN$ |
| Relative Change from Baseline | | Decrease ≥ 20 and < LLN |

To identify LVEF values of potential clinical importance, NCI-CTCAE v4.0 will be used to assign categories that align with the grades for 'Ejection fraction decreased'.

# 13.9. Appendix 9: Population Pharmacokinetic (PopPK) Analyses

Not applicable.

201973

# 13.10. Appendix 10: Abbreviations & Trademarks

# 13.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| AI | Aromatase Inhibitor |
| ALT | Alanine Aminotransferase |
| AST | Aspartate Aminotransferase |
| ATC | Anatomical-Therapeutic-Chemical |
| BOR | Best Overall Response |
| BP | Blood Pressure |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling and Simulation |
| CR | Complete Response |
| CSR | Clinical Study Report |
| | , 1 |
| CY | Common Terminology Criteria for Adverse Events |
| eCRF | Electronic Case Report Form |
| EORTC-QLQ-C30 | European Organization for Research and Treatment of Cancer Quality |
| EORTC-QLQ-BR23 | European Organization for Research and Treatment of Cancer Quality |
| EudraCT | European Union Drug Regulating Authorities Clinical Trials Database |
| HLGT | High Level Group Term |
| HR+/HER2-BC | Hormone Receptor-Positive/HER2-Negative Breast Cancer |
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| IDSL | Integrated Data Standards Library |
| IM | Intramuscular(ly) |
| INR | International Normalized Ratio |
| LLN | Lower Limit of Normal |
| | Left Ventricular Ejection Fraction |
| | 5 |
| EORTC-QLQ-BR23 EudraCT HLGT HR+/HER2- BC IA ICH IDSL IM INR | of Life Questionnaire Core-30 European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Breast-23 European Union Drug Regulating Authorities Clinical Trials Database High Level Group Term Hormone Receptor-Positive/HER2-Negative Breast Cancer Interim Analysis International Conference on Harmonisation Integrated Data Standards Library Intramuscular(ly) International Normalized Ratio Lower Limit of Normal |

201973

| Abbreviation | Description |
|--------------|----------------------------------------------------------|
| MUGA | Multiple Gated Acquisition |
| NCI | National Cancer Institute |
| NE | Not Evaluable |
| ORR | Objective Response Rate |
| OS | Overall Survival |
| PD | Progressive Disease |
| PFS | Progression-Free Survival |
| PK | Pharmacokinetic |
| PR | Partial Response or ECG parameter (context dependent) |
| PRO | Patient Reported Outcomes |
| PT | Preferred Term |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| RAP | Reporting and Analysis Plan |
| RECIST | Response Evaluation Criteria in Solid Tumors |
| RP2D | Recommended Phase 2 Dose |
| RS | Response Dataset |
| RUCAM | Roussel Uclaf Causality Assessment Method |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SD | Standard Deviation or Stable Disease (context dependent) |
| SDTM | Study Data Tabulation Model |
| SMQ | Standardised MedDRA Query |
| SOC | System Organ Class |
| SOP | Standard Operation Procedure |
| TEAE | Treatment-Emergent Adverse Event |
| TFL | Tables, Figures, and Listings |
| ULN | Upper Limit of Normal |

# 13.10.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies | Trademarks not owned by the GlaxoSmithKline Group of Companies |
|---|---|
| None | SAS |

201973

# 13.11. Appendix 11: List of Data Displays

# 13.11.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|------------|
| Study Population | 1.1 to 1.22 | N.A. |
| Efficacy | 2.1 to 2.3 | 2.1 to 2.3 |
| Safety | 3.1 to 3.51 | N.A. |
| Pharmacokinetic | 4.1 to 4.8 | 4.1 to 4.5 |
| Section | Listings | |
| ICH Listings | 1 to 50 | |
| Other Listings | 51 to 71 | |

# 13.11.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 12: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |

**NOTES:** Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 13.11.3. Deliverables

| Delivery | Description |
|----------|-------------------------------------------------|
| IA | Interim Analysis |
| RP2D | Recommended Phase 2 Dose Analysis |
| SAC | Final Statistical Analysis Complete for Phase I |

201973

# 13.11.4. Study Population Tables

| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Subjec | t Disposition | | | | |
| 1.1. | All Treated | ES1 | Summary of Subject Status and Reason for Study<br>Withdrawal | | RP2D, SAC |
| 1.2. | All<br>Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | | SAC |
| 1.3. | All Treated | SD4 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | Order the Reasons as displayed in the eCRF; present treatment status and reasons separately for GSK525762, fulvestrant, and overall within the same table. | IA, RP2D, SAC |
| Popula | Populations Analysed | | | | |
| 1.4. | All<br>Screened | SP1 | Summary of Study Population | | IA, RP2D, SAC |
| Protoc | Protocol Deviations | | | | |

201973

| 1.5. | All Treated | DV1 | Summary of Major Protocol Deviations | | RP2D, SAC |
|---|---|---|---|---|---|
| Demog | raphic and Ba | seline Chara | acteristics | | |
| 1.6. | All Treated | DM1 | Summary of Demographic Characteristics | | IA, RP2D, SAC |
| 1.7. | All Treated | DM6 | Summary of Race and Racial Combinations | | RP2D, SAC |
| 1.8. | All Treated | DM11 | Summary of Age Ranges | | RP2D, SAC |
| 1.9. | All Treated | PS1A | Summary of ECOG Performance Status at Baseline | Only include baseline visit from standard. | RP2D, SAC |
| 1.10. | All Treated | LA1 | Summary of Disease Burden at Baseline | | RP2D, SAC |
| 1.11. | All Treated | DC1 | Summary of Disease Characteristics at Initial Diagnosis | | IA, RP2D, SAC |
| 1.12. | All Treated | DC2 | Summary of Disease Characteristics at Screening | | IA, RP2D, SAC |
| 1.13. | All Treated | MD1 | Summary of Metastatic Disease at Screening | | RP2D, SAC |
| Prior a | nd Concomita | nt Medication | ons | | |
| 1.14. | All Treated | MH1 | Summary of Past Medical Conditions | | RP2D, SAC |
| 1.15. | All Treated | MH1 | Summary of Current Medical Conditions | | RP2D, SAC |
| 1.16. | All Treated | OSP1 | Summary of Prior Cancer-Related Surgical Procedures | | RP2D, SAC |
| 1.17. | All Treated | OSP1 | Summary of On-Treatment Cancer-Related Surgical Procedures | | RP2D, SAC |

201973

| 1.18. | All Treated | CM8 | Summary of Concomitant Medication by Ingredient | Medications to be sorted in descending order of overall incidence. | RP2D, SAC |
|---|---|---|---|---|---|
| Anti-Ca | ancer Therapi | es | | | |
| 1.19. | All Treated | AC1 | Summary of Prior Anti-Cancer Therapy | Present all therapies (including radiotherapies). | IA, RP2D, SAC |
| 1.20. | All Treated | CM1 | Summary of Prior Dictionary Coded Anti-Cancer<br>Therapy | | RP2D, SAC |
| 1.21. | All Treated | AC3 | Summary of Number of Anti-Cancer Therapy<br>Regimens | | RP2D, SAC |
| 1.22. | All Treated | AC4 | Summary of Best Response to Prior Anti-Cancer<br>Therapy | | RP2D, SAC |

# 13.11.5. Efficacy Tables

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Overal | Overall Response Rate | | | | |

201973

| 2.1. | Modified All<br>Treated | RE1a | Summary of Investigator Assessed Best<br>Response (RECIST v1.1 Criteria) | Show all categories of BOR, including CR and PR each split up into confirmed and unconfirmed. Categories would then include: CR confirmed, CR, unconfirmed, PR confirmed, PR unconfirmed, SD, PD, and NE. Also, include ORR and DCR (as defined in this RAP). | IA, SAC |
|---|---|---|---|---|---|
| Second | lary Endpoints | | | | |
| 2.2. | Modified All<br>Treated | TTE6 | Summary of Duration of Response | | RP2D, SAC |
| 2.3. | Modified All<br>Treated | TTE6 | Summary of Progression-Free Survival | Produce only if data warrant. | RP2D, SAC |

# 13.11.6. Efficacy Figures

| Efficacy: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID | Title | Programming Notes | Deliverable |
| | | / Example Shell | | | [Priority] |
| 2.1. | Modified | RE8A | Waterfall Plot of Maximum Percent Reduction | The plot will be color-coded for | IA, RP2D, |
| | All Treated | | from Baseline in Tumour Measurement (Target | best overall response with | SAC |
| | | | Lesions) | confirmation. Indication of the | |
| | | | , | subject number and dose and | |
| | | | | cohort will be provided below the | |

201973

| | | | | plot. Max percent reduction will be based on target lesions. | |
|---|---|---|---|---|---|
| 2.2. | Modified<br>All Treated | Non-Standard 1 | Spider Plot of Percent Change from Baseline in<br>Target Lesion Diameter | | IA, RP2D,<br>SAC |
| 2.3. | Modified<br>All Treated | TTE10 | Kaplan-Meier Plot of Progression-Free Survival | | RP2D, SAC |

# 13.11.7. Safety Tables

| Safety | Safety: Tables | | | | | | |
|---|---|---|---|---|---|--|--|
| No. | Population | IDSL / TST ID<br>/ Example Shell | Title | Programming Notes | Deliverable<br>[Priority] | | |
| Expos | ure | | | , | | | |
| 3.1. | All Treated | OEX1 | Summary of Exposure to GSK525762 | In OEX1, the time on study treatment categories can be modified if necessary. | IA, RP2D, SAC | | |
| 3.2. | All Treated | OEX5 | Summary of Exposure to Fulvestrant | In OEX5, the categories of number of subjects who received a given number of cycles can be modified if necessary. | IA, RP2D, SAC | | |
| 3.3. | All Treated | ODMOD1 | Summary of Dose Delays/Interruptions of GSK525762 | This may be replaced by a listing if minimal data available. | RP2D, SAC | | |
| 3.4. | All Treated | ODMOD1 | Summary of Dose Reductions of GSK525762 | This may be replaced by a listing if minimal data available. | RP2D, SAC |
|---|---|---|---|---|---|
| 3.5. | All Treated | ODMOD8 | Summary of Dose Escalations of GSK525762 | This may be replaced by a listing if minimal data available. | RP2D, SAC |
| 3.6. | All Treated | ODMOD3 | Summary of Dose Delays/Interruptions of Fulvestrant | | RP2D, SAC |
| 3.7. | All Treated | ODMOD1 | Summary of Dose Reductions of Fulvestrant | | RP2D, SAC |
| 3.8. | All Treated | ODMOD4 | Summary of Missed Doses of Fulvestrant | | RP2D, SAC |
| 3.9. | All Treated | AE19 | Summary of Dose-Limiting Toxicities during the Determinative Period | | RP2D, SAC |
| Adver | se Events | | | | L |
| 3.10. | All Treated | AE13 | Adverse Event Overview | | IA, SAC |
| 3.11. | All Treated | AE16 | Summary of All Adverse Events by System<br>Organ Class and Preferred Term | | RP2D, SAC |
| 3.12. | All Treated | AE5B | Summary of Adverse Events of Special Interest<br>Regardless of Relatedness | | IA, RP2D, SAC |
| 3.13. | All Treated | AE5B | Summary of Adverse Events of Special Interest<br>by Maximum Grade Regardless of Relatedness | | RP2D, SAC |

| 3.14. | All Treated | AE5B | Summary of Drug-Related Adverse Events by<br>System Organ Class and Preferred Term and<br>Maximum Grade | Include Any Treatment-Related, GSK525762-Related, and Fulvestrant-Related in the same table, with separate headers and starting on separate pages. | RP2D, SAC |
|---|---|---|---|---|---|
| 3.15. | All Treated | AE5B | Summary of All Adverse Events by System<br>Organ Class and Preferred Term and<br>Maximum Grade | | IA, RP2D, SAC |
| 3.16. | All Treated | AE13 | Summary of Grade 3-4 Adverse Events<br>Overview | | RP2D, SAC |
| 3.17. | All Treated | AE3 | Summary of Drug-Related Adverse Events by Maximum Grade 3-4 | Include Total Column. Include Any Treatment-Related, GSK525762-Related, and Fulvestrant-Related in the same table, with separate headers and starting on separate pages. | RP2D, SAC |
| 3.18. | All Treated | AE3 | Summary of Adverse Events Leading to<br>Permanent Discontinuation of Study Treatment | Include Any Treatment,<br>GSK525762, and Fulvestrant in the<br>same table, with separate headers<br>and starting on separate pages. | IA, RP2D, SAC |
| 3.19. | All Treated | AE3 | Summary of Adverse Events Leading to Dose<br>Reductions in Study Treatment | Include Any Treatment,<br>GSK525762, and Fulvestrant in the<br>same table, with separate headers<br>and starting on separate pages. | IA, RP2D, SAC |

| 3.20. | All Treated | AE3 | Summary of Adverse Events Leading to Dose<br>Delays or Interruptions in Study Treatment | Include Any Treatment,<br>GSK525762, and Fulvestrant in the<br>same table, with separate headers<br>and starting on separate pages. | IA, RP2D, SAC |
|---|---|---|---|---|---|
| 3.21. | All Treated | AE15 | Summary of Common (>=5%) Non-serious<br>Adverse Events by System Organ Class and<br>Preferred Term (Number of Subjects and<br>Occurrences) | | RP2D, SAC |
| 3.22. | All Treated | AE16 | Summary of Serious Adverse Events by<br>System Organ Class and Preferred Term<br>(Number of Subjects and Occurrences) | | RP2D, SAC |
| 3.23. | All Treated | AE3 | Summary of Drug-Related Serious Adverse<br>Events | Include Any Treatment-Related, GSK525762-Related, and Fulvestrant-Related in the same table. Page by these categories with header description in top left-hand corner. | IA, RP2D, SAC |
| 3.24. | All Treated | AE20 | Summary of Drug-Related Non-Fatal Serious<br>Adverse Events | Include Any Treatment-Related, GSK525762-Related, and Fulvestrant-Related in the same table. Page by these categories with header description in top left-hand corner. | RP2D, SAC |
| 3.25. | All Treated | AE3 | Summary of Adverse Events Classified as Dose-Limiting Toxicities (DLTs) | | RP2D, SAC |

| 3.26. | All Treated | ESI1 | Summary of Characteristics of Adverse Events of Special Interest | This table will be presented individually for each category of AESI. | SAC |
|---|---|---|---|---|---|
| 3.27. | All Treated | ESI2b | Summary of Onset and Duration of the First<br>Occurrence of Adverse Events of Special<br>Interest | This table will be presented individually for each category of AESI. | SAC |
| 3.28. | All Treated | DD1 | Summary of Deaths | | RP2D, SAC |
| Labor | atory: Chemi | stry | | | |
| 3.29. | All Treated | LB1 | Summary of Chemistry Changes from Baseline | | SAC |
| 3.30. | All Treated | LB18 | Summary of Chemistry Grade Changes from Baseline | For lab tests that are graded, include worst-case changes. | RP2D, SAC |
| 3.31. | All Treated | LB3 | Summary of Chemistry Changes from Baseline with Respect to the Normal Range | For lab tests that are graded, include worst-case changes. | RP2D, SAC |
| Labor | atory: Haema | tology | | | |
| 3.32. | All Treated | LB1 | Summary of Haematology Changes from Baseline | | SAC |
| 3.33. | All Treated | LB18 | Summary of Haematology Grade Changes from Baseline | For lab tests that are graded. | RP2D, SAC |
| 3.34. | All Treated | LB3 | Summary of Haematology Changes from<br>Baseline with Respect to the Normal Range | For lab tests that are graded. | RP2D, SAC |

| Labor | Laboratory: Liver Events | | | | |
|---|---|---|---|---|---|
| 3.35. | All Treated | LIVER1 | Summary of Liver Monitoring/Stopping Event<br>Reporting | | SAC |
| 3.36. | All Treated | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities Including Possible Hy's Law Cases | Summarize by ascending dose level and total. Possible Hy's law cases will be defined as any event of either: (a) ALT ≥3 × the upper limit of normal (ULN) and bilirubin ≥2 × ULN (>35% direct bilirubin) or (b) ALT ≥3 × ULN and INR >1.5, if INR is measured. Total bilirubin ≥2 × ULN can be within 28 days following the ALT elevation and, if direct bilirubin is available on the same day, it must be ≥35% of total bilirubin. | SAC |

| Urinal | ysis | | | | |
|---|---|---|---|---|---|
| 3.37. | All Treated | UR1 | Summary of Worst-Case Urinalysis Result<br>Increases from Baseline | Include tests done by Dipstick –<br>Specific gravity, pH, Glucose,<br>Protein, Blood, Ketones. | RP2D, SAC |
| 3.38. | All Treated | LB18 | Summary of Urinalysis Grade Changes from Baseline | For lab tests that are graded. | RP2D, SAC |
| Coagu | Coagulation | | | | |
| 3.39. | All Treated | LB3 | Summary of Coagulation Changes from<br>Baseline with Respect to Normal Range | | SAC |

| Vital S | Vital Signs | | | | |
|---|---|---|---|---|---|
| 3.40. | All Treated | VS1 | Summary of Vital Signs | Include all parameters (heart rate, diastolic blood pressure, systolic blood pressure, respiratory rate, and temperature). | RP2D, SAC |
| 3.41. | All Treated | VS1 | Summary of Vital Sign Changes from Baseline | Again, show changes from baseline for all parameters (heart rate, diastolic blood pressure, systolic blood pressure, respiratory rate, and temperature). | RP2D, SAC |
| ECG | | | | | |

| 3.42. | All Treated | EG1 | Summary of ECG Findings | | RP2D, SAC |
|---|---|---|---|---|---|
| 3.43. | All Treated | EG2 | Summary of Change from Baseline in ECG<br>Values | | RP2D, SAC |
| 3.44. | All Treated | EG10A | Summary of Maximum QTcF Value Post-Baseline Relative to Baseline | Include QTcF > 500 msec. Include footnote for baseline definition. Specify the data source in the title (i.e., local read vs. central read). Also, add footnote: "Only the post-baseline assessments that used the same source as the baseline assessment (i.e., local or central cardiologist read) are used to derive change from baseline." | RP2D, SAC |
| 3.45. | All Treated | EG11A | Summary of Maximum Increase in QTcF<br>Values Post-Baseline Relative to Baseline | Include QTcF > 500 msec. Include footnote for baseline definition. Specify the data source in the title (i.e., local read vs. central read). Also, add footnote: "Only the post-baseline assessments that used the same source as the baseline assessment (i.e., local or central | RP2D, SAC |

| | | | | cardiologist read) are used to derive change from baseline." | |
|---|---|---|---|---|---|
| Perfor | mance Status | | | | |
| 3.46. | All treated | PS1A | Summary of ECOG Performance Status | | RP2D, SAC |
| 3.47. | All treated | PS3A | Summary of Change in ECOG Performance<br>Status from Baseline | | RP2D, SAC |
| Left V | entricular Ej | ection Fraction | | 1 | |
| 3.48. | All Treated | OLVEF1A | Summary of Change from Baseline in Left<br>Ventricular Ejection Fraction | | RP2D, SAC |
| Value | Evidence and | Outcomes | | | |
| 3.49. | All Treated | SF4_NS2 | Summary of and Change from Baseline in EORTC-QLQ-C30 | | SAC |
| 3.50. | All Treated | SF4_NS2 | Summary of and Change from Baseline in QLQ-BR23 | | SAC |
| 3.51. | All Treated | SF4_NS2 | Summary of and Change from Baseline in PRO-CTCAE | | SAC |

201973

### 13.11.8. Pharmacokinetic Tables

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Drug | Concentration | 1 Measure | | | |
| 4.1. | PK | PK01 | Summary of GSK525762 Pharmacokinetic<br>Concentration-Time Data by Dose Level and<br>Cohort | Use descriptive statistics (n, mean, SD, median, min and max) by planned relative assessment time; concentrations in ng/mL | RP2D, SAC |
| 4.2. | PK | PK01 | Summary of GSK3529246 Pharmacokinetic<br>Concentration-Time Data by Dose Level and<br>Cohort | Use descriptive statistics (n, mean, SD, median, min and max) by planned relative assessment time; concentrations in ng/mL | RP2D, SAC |
| 4.3. | PK | PK01 | Summary of Total Active Moiety of GSK525762<br>Pharmacokinetic Concentration-Time Data by<br>Dose Level and Cohort | Use descriptive statistics (n, mean, SD, median, min and max) by planned relative assessment time; TAM concentration in nM | RP2D, SAC |
| 4.4. | PK | PK01 | Summary of Fulvestrant Pharmacokinetic<br>Concentration-Time Data by Dose Level and<br>Cohort | Summary presented only for predose as fulvestrant samples are collected only at pre-dose; use descriptive statistics (n, mean, SD, median, min and max) by planned relative assessment time; concentrations in ng/mL | RP2D, SAC |

| Pharn | Pharmacokinetic Parameters | | | | |
|---|---|---|---|---|---|
| 4.5. | PK | PK06 | Summary of Derived GSK525762 Pharmacokinetic Parameters | PK parameters: C <sub>max</sub> , T <sub>max</sub> , C <sub>trough</sub> determined from the concentration-time data in ng/ml and in nM after conversion from ng/mL to nM; descriptive summaries: mean, SD, median, min, max, geometric mean & SD, CV%, and 95%CI of log-transformed parameters, if applicable | RP2D, SAC |
| 4.6. | PK | PK06 | Summary of Derived GSK3529246 Pharmacokinetic Parameters | PK parameters: C <sub>max</sub> , T <sub>max</sub> , C <sub>trough</sub> determined from the concentration-time data in ng/ml and in nM after conversion from ng/mL to nM; descriptive summaries: mean, SD, median, min, max, geometric mean & SD, CV%, and 95%CI of log-transformed parameters, if applicable | RP2D, SAC |
| 4.7. | PK | PK06 | Summary of Derived Total Active Moiety of GSK525762 Pharmacokinetic Parameters | PK parameters: C <sub>max</sub> , T <sub>max</sub> , C <sub>trough</sub> determined from the concentration-time data after conversion from ng/mL to nM; descriptive summaries: mean, SD, median, min, max, geometric mean & SD, CV%, and 95%CI of log-transformed parameters, if applicable | SAC |

201973

| 4.8. | PK | PK06 | Summary of Derived Fulvestrant Pharmacokinetic Parameters | PK parameters: C <sub>max</sub> , T <sub>max</sub> , C <sub>trough</sub> determined from the concentration-time data in ng/ml and in nM after conversion from ng/mL to nM; descriptive summaries: mean, SD, median, min, max, geometric mean & SD, CV%, and 95%CI of log-transformed parameters, if applicable | RP2D, SAC |
|---|---|---|---|---|---|
|---|---|---|---|---|---|

## 13.11.9. Pharmacokinetic figures

| Pharmacokinetic: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Drug | Concentration | Measure | | | |
| 4.1. | PK | PK17 | Overlay of Mean GSK525762 (nM), Mean GSK3529246 (nM), and Mean Total Active Moiety of GSK525762 (nM) Concentration-Time Curves | Include both Wk1 and Wk3 (on separate plots within the panel) and, for each, show both linear and semi-log curves. | SAC |
| 4.2. | PK | PK18 | Overlay of Median GSK525762 (nM), Median GSK3529246 (nM), and Median Total Active Moiety of GSK525762 (nM) Concentration-Time Curves | Include both Wk1 and Wk3 (on separate plots within the panel) and, for each, show both linear and semi-log curves. | SAC |

201973

| 4.3. | PK | PK16 | GSK525762 (ng/mL) Concentration-Time Curves by Dose Level/Cohort and Week | Overlay the curves for the different dose level/cohorts on the same plot but show separate plots within the panel for Wk 1 and Wk 3; concentration in ng/mL. | SAC |
|---|---|---|---|---|---|
| 4.4. | PK | PK16 | GSK3529246 (ng/mL) Concentration-Time Curves by Dose Level/Cohort and Week | Overlay the curves for the different dose level/cohorts on the same plot but show separate plots within the panel for Wk 1 and Wk 3; concentration in ng/mL. | SAC |
| 4.5. | PK | PK16 | Total Active Moiety of GSK525762 (nM) Concentration-Time Curves by Dose Level/Cohort and Week | Overlay the curves for the different dose level/cohorts on the same plot but show separate plots within the panel for Wk 1 and Wk 3; concentration in nM. | SAC |

# 13.11.10. ICH Listings

| ICH: I | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | Subject Disposition | | | | |

| 1. | All Treated | ES2 | Listing of Reasons for Subject Withdrawal | RP2D, SAC |
|---|---|---|---|---|
| 2. | All Screened | ES7 | Listing of Reasons for Screen Failure | SAC |
| 3. | All Treated | SD2 | Listing of Reasons for Study Treatment Discontinuation | RP2D, SAC |
| Popula | Populations Analysed | | | |
| 4. | All Screened | SP3 | Listing of Subjects Excluded from Any population | RP2D, SAC |

| Proto | ocol Deviations | | | |
|---|---|---|---|---|
| 5. | All Treated | DV2 | Listing of Protocol Deviations | RP2D, SAC |
| 6. | All Treated | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | SAC |
| Basel | ine and Disease | Characteristics | | |
| 7. | All Treated | DM2 | Listing of Demographic Characteristics | RP2D, SAC |
| 8. | All Treated | DM9 | Listing of Race | RP2D, SAC |
| Treat | tment Exposure | | | |
| 9. | All Treated | TA1 | Listing of Planned and Actual Treatments | RP2D, SAC |
| 10. | All Treated | COMP3C | Listing of GSK525762 Drug Accountability | RP2D, SAC |

| 11. | All Treated | OEX3a | Listing of Exposure Data to GSK525762 | RP2D, SAC |
|---|---|---|---|---|
| 12. | All Treated | OEX8B | Listing of Exposure Data to Fulvestrant | RP2D, SAC |
| 13. | All Treated | ODMOD10A | Listing of Dose Reductions for GSK525762 | RP2D, SAC |
| 14. | All Treated | ODMOD10A | Listing of Dose Reductions for Fulvestrant | SAC |
| 15. | All Treated | ODMOD11A | Listing of Dose Interruptions/Delays for GSK525762 | RP2D, SAC |
| 16. | All Treated | ODMOD11A | Listing of Dose Interruptions/Delays for Fulvestrant | RP2D, SAC |
| 17. | All Treated | ODMOD11A | Listing of Missed Doses for Fulvestrant | RP2D, SAC |
| 18. | All Treated | ODMOD15A | Listing of Dose Escalations for GSK525762 | RP2D, SAC |
| Adver | se Events | | | |
| 19. | All Treated | OAE04 | Listing of All Adverse Events | RP2D, SAC |
| 20. | All Treated | OAE03 | Listing of Subject Numbers for Individual Adverse<br>Events | RP2D, SAC |
| 21. | All Treated | OAE04 | Listing of Dose-Limiting Adverse Events | RP2D, SAC |
| 22. | All Treated | AE2 | Listing of Relationship Between Adverse Event System<br>Organ Class, Preferred Term and Verbatim Text | SAC |
| Seriou | s and Other Sig | nificant Adverse | Events | , |
| 23. | All Treated | OAE04 | Listing of Fatal Serious Adverse Events | RP2D, SAC |

| 24. | All Treated | OAE04 | Listing of Non-Fatal Serious Adverse Events | | RP2D, SAC |
|---|---|---|---|---|---|
| 25. | All Treated | OAE04 | Listing of Adverse Events Leading to Permanent<br>Discontinuation of Study Treatment | Based on Action taken question on AE/SAE. | RP2D, SAC |
| 26. | All Treated | OAE04 | Listing of Adverse Events Leading to Dose Reductions for any Study Drug | | RP2D, SAC |
| 27. | All Treated | OAE04 | Listing of Adverse Events Leading to Dose<br>Interruptions/Delays for any Study Drug | | RP2D, SAC |
| 28. | All Treated | AE14 | Listing of Reasons for Considering as a Serious Adverse<br>Event | | SAC |
| 29. | All Treated | OAE04 | Listing of Adverse Events of Special Interest | | SAC |
| Dose- | Limiting Toxici | ty | | | |
| 30. | All Treated | DL3 | Listing of Dose-Limiting Toxicities during the Determinative Period | | RP2D, SAC |
| Labo | ratory | | | 1 | |
| 31. | All Treated | LB13 | Listing of Chemistry Laboratory Data for Subjects with Lab Values Outside of Normal Range | | SAC |
| 32. | All Treated | LB13 | Listing of Haematology Laboratory Data for Subjects with Lab Values Outside of Normal Range | | SAC |
| 33. | All Treated | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | | SAC |

| 34. | All Treated | LIVER13 | Listing of Subjects Meeting Hepatobiliary Laboratory<br>Criteria Post-Baseline | | SAC |
|---|---|---|---|---|---|
| 35. | All Treated | UR2A | Listing of Urinalysis Data for Subjects with Any Value of Potential Clinical Importance | | RP2D, SAC |
| 36. | All Treated | LB13 | Listing of Coagulation and Other Laboratory data | | SAC |
| 37. | All Treated | OLB7 | Listing of Coagulation and Other Laboratory Data for<br>Subjects with Lab Values Outside of Normal Range | | SAC |
| 38. | All Treated | LB14 | Listing of Laboratory Data with Character Results | | SAC |
| Pharm | nacokinetic | | | | |
| 39. | PK | PK07 | Listing of GSK525762 Pharmacokinetic Concentration-<br>Time Data by dose level and population | In ng/mL and nM. | RP2D, SAC |
| 40. | PK | PK07 | Listing of GSK3529246 Pharmacokinetic<br>Concentration-Time Data by dose level and population | In ng/mL and nM. | SAC |
| 41. | PK | PK07 | Listing of Total Active Moiety of GSK525762 Pharmacokinetic Concentration-Time Data by dose level and population | In nM. | SAC |
| 42. | PK | PK07 | Listing of Fulvestrant Pharmacokinetic Concentration-<br>Time Data by dose level and population | In ng/mL. | SAC |
| 43. | PK | PK13 | Listing of Derived GSK525762 (nM) Pharmacokinetic Parameters | C <sub>max</sub> , T <sub>max</sub> , C <sub>trough</sub> , determined from | RP2D, SAC |

| | | | | concentration (ng/mL) - time data. | |
|---|---|---|---|---|---|
| 44. | PK | PK13 | Listing of Derived GSK3529246 (nM) Pharmacokinetic Parameters | C <sub>max</sub> , T <sub>max</sub> , C <sub>trough</sub> ,<br>determined from<br>concentration (ng/mL) -<br>time data. | SAC |
| 45. | PK | PK13 | Listing of Derived Total Active Moiety of GSK525762 (nM) Pharmacokinetic Parameters | C <sub>max</sub> , T <sub>max</sub> , C <sub>trough</sub> ,<br>determined from<br>concentration (nM) - time<br>data. | SAC |
| Effica | ncy | <u>I</u> | | | |
| 46. | All Evaluable | RE12 | Listing of Subject Best Response for Interim Review by First Dose Date | Sort by date of first dose. | IA |
| 47. | Modified All<br>Treated | LA2 | Listing of Investigator-Assessed Target Lesions (RECIST v1.1 Criteria) | | RP2D, SAC |
| 48. | Modified All<br>Treated | LA3 | Listing of Investigator-Assessed Non-Target Lesions (RECIST v1.1 Criteria) | | RP2D, SAC |
| 49. | Modified All<br>Treated | LA4 | Listing of Investigator-Assessed New Lesions (RECIST v1.1 Criteria) | | RP2D, SAC |
| 50. | Modified All<br>Treated | RE5 | Listing of Investigator-Assessed Best Overall Responses (RECIST v1.1) | | RP2D, SAC |

201973

# 13.11.11. Non-ICH Listings

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Demo | graphic and B | Baseline Characteris | stics | | |
| 51. | All Treated | SU2 | Listing of Substance Use | | SAC |
| 52. | All Treated | DC3 | Listing of Disease Characteristics at Initial Diagnosis | | RP2D, SAC |
| 53. | All Treated | DC4 | Listing of Disease Characteristics at Screening | | RP2D, SAC |
| 54. | All Treated | MD2 | Listing of Metastatic Disease at Screening | | RP2D, SAC |
| Prior | and Concomit | tant Medication | | | <u> </u> |
| 55. | All Treated | МН2 | Listing of Medical Conditions | Include Prior and Current, with Status column indicating same. | RP2D, SAC |
| 56. | All Treated | CM2 | Listing of Concomitant Medications | | SAC |
| 57. | All Treated | BP4 | Listing of Blood Products or Blood Supportive Care<br>Products | Include Prior (BP4) and On-<br>Treatment (BP5). | SAC |
| 58. | All Treated | OSP3 | Listing of Surgical Procedures | Include Prior and On-<br>Treatment. | SAC |

| 59. | All Treated | AE2 | Listing of Relationship Between ATC Level1,<br>Ingredient and Verbatim Text | | SAC |
|---|---|---|---|---|---|
| Anti- | Anti-Cancer Therapy | | | | |
| 60. | All Treated | AC6 | Listing of All Anti-Cancer Therapy | Including Prior and Subsequent. | RP2D, SAC |
| 61. | All Treated | AC7 | Listing of Anti-Cancer Radiotherapy | Including Prior and Subsequent. | RP2D, SAC |
| ECG | | | | 1 | |
| 62. | All Treated | EG5 | Listing of All ECG Findings for Subjects with an Abnormal Finding | | RP2D, SAC |
| 63. | All Treated | EG3 | Listing of ECG Values for Subjects with Abnormal Values | | RP2D, SAC |
| 64. | All Treated | EG3 | Listing of QTcF Values of Potential Clinical Importance | | SAC |
| Vital | Signs | l | | | |
| 65. | All Treated | VS4 | Listing of Vital Signs | | SAC |
| 66. | All Treated | OVT7A | Listing of Vital Signs with Abnormal Values | | RP2D, SAC |
| LVEF | 7 | | | | |
| 67. | All Treated | OLVEF2A | Listing of Left Ventricular Ejection Fraction Results | | RP2D, SAC |
| Labor | Laboratory | | | | |

| 68. | All Treated | OLB13 | Listing of Laboratory Data with Character Results | SAC |
|---|---|---|---|---|
| Value | Value Evidence and Outcomes | | | |
| 69. | Modified<br>All Treated | SF6 | Listing of EORTC-QLQ-C30 Results | SAC |
| 70. | Modified<br>All Treated | SF6 | Listing of EORTC-QLQ-BR23 Results | SAC |
| 71. | Modified<br>All Treated | SF6 | Listing of PRO-CTCAE Results | SAC |

201973

### 13.12. Appendix 12: Example Mock Shells for Data Displays

Example Non-Standard 1

Protocol: 201973

Page 1 of 1 Population: Modified All Treated (Data as of: 30MAY2013)

Figure 1 Spider Plot of Percent Change from Baseline In Target Lesion Diameter

